#### TITLE PAGE

**PROTOCOL TITLE:** A Multicenter, Randomized, Double-Blind,

Placebo-Controlled, Multiple Dose Study to Evaluate the

Efficacy and Safety of VIS649 in Participants with

Immunoglobulin A (IgA) Nephropathy

PROTOCOL NUMBER: VIS649-201

COMPOUND VIS649

STUDY PHASE Phase 2

**SHORT TITLE:** Phase 2 Study of VIS649 for IgA Nephropathy

VERSION: 2.0

**VERSION DATE:** 01 November 2019

**SPONSOR:** Visterra, Inc.

275 2<sup>nd</sup> Avenue

Waltham, MA 02451

#### **REGULATORY AGENCY IDENTIFIER NUMBER(S)**

**IND Number:** 135,282

NCT TBD

**EudraCT Number:** 2019-002531-29

# **APPROVAL PAGE**

**PROTOCOL TITLE:** A Multicenter, Randomized, Double-Blind, Placebo-Controlled,

Multiple Dose Study to Evaluate the Efficacy and Safety of

VIS649 in Participants with Immunoglobulin A (IgA) Nephropathy

This Clinical Study Protocol has been reviewed and approved by the Sponsor in order to ensure compliance with Good Clinical Practice.

#### **Sponsor Signatory:**



### TABLE OF CONTENTS

| 1. | PROTOCOL SUMMARY | 7 |
|-------|-------------------------------------------------------|----|
| 1.1 | Synopsis | 7 |
| 1.2 | Schema | 16 |
| 1.3 | Schedule of Assessments | 17 |
| 2. | INTRODUCTION | 20 |
| 2.1 | Study Rationale | 20 |
| 2.2 | Background | 21 |
| 2.3 | Benefit/Risk Assessment | 23 |
| 2.3.1 | Risk Assessment | 23 |
| 2.3.2 | Benefit Assessment | 26 |
| 2.3.3 | Overall Benefit: Risk Conclusion | 26 |
| 3. | OBJECTIVES AND ENDPOINTS | 28 |
| 4. | STUDY DESIGN | 31 |
| 4.1 | Overall Design | 31 |
| 4.2 | Scientific Rationale for Study Design | 33 |
| 4.3 | Justification for Dose | 35 |
| 4.4 | End of Study Definition | 36 |
| 5. | STUDY POPULATION | 37 |
| 5.1 | Inclusion Criteria | 37 |
| 5.2 | Exclusion Criteria | 38 |
| 5.3 | Lifestyle Considerations | 40 |
| 5.4 | Screen Failures | 40 |
| 6. | STUDY INTERVENTION | 41 |
| 6.1 | Study Intervention(s) Administered | 41 |
| 6.2 | Preparation/Handling/Storage/Accountability | 42 |
| 6.3 | Measures to Minimize Bias: Randomization and Blinding | 42 |
| 6.4 | Study Intervention Compliance | 43 |
| 6.5 | Concomitant Therapy | 43 |
| 6.5.1 | Concomitant Therapy to be Avoided | 43 |

| 6.6 | Dose Modification | 44 |
|---|---|---|
| 6.7 | Intervention after the End of the Study | 44 |
| 7. | DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL | 45 |
| 7.1 | Discontinuation of Study Intervention Dosing | 45 |
| 7.1.1 | Temporary Discontinuation | 45 |
| 7.1.2 | Rechallenge | 45 |
| 7.2 | Participant Discontinuation/Withdrawal from the Study | 46 |
| 7.3 | Lost to Follow-up | 46 |
| 8. | STUDY ASSESSMENTS AND PROCEDURES | 47 |
| 8.1 | Efficacy Assessments | 47 |
| 8.1.1 | Twenty-four-hour Urine Sample Collection | 47 |
| 8.2 | Safety Assessments | 47 |
| 8.2.1 | Physical Examinations | 47 |
| 8.2.2 | Vital Signs | 47 |
| 8.2.3 | Electrocardiograms | |
| 8.2.4 | Clinical Safety Laboratory Assessments | 48 |
| 8.3 | Adverse Events and Serious Adverse Events | |
| 8.3.1 | Time Period and Frequency for Collecting Adverse Event and Serious Adverse Event Information | 49 |
| 8.3.2 | Method of Detecting Adverse Events and Serious Adverse Events | 49 |
| 8.3.3 | Follow-up of Adverse Events and Serious Adverse Events | 50 |
| 8.3.4 | Regulatory Reporting Requirements for Serious Adverse Events | 50 |
| 8.3.5 | Pregnancy | 51 |
| 8.4 | Treatment of Overdose | 51 |
| 8.5 | Pharmacokinetics | 51 |
| 8.6 | Pharmacodynamics | 52 |
| 8.7 | Genetics | 52 |
| 8.8 | Biomarkers | 52 |
| 8.9 | Immunogenicity Assessments | 53 |
| 8.10 | Medical Resource Utilization and Health Economics | 53 |


| 9. | STATISTICAL CONSIDERATIONS | 54 |
|---|---|---|
| 9.1 | Statistical Hypothesis | 54 |
| 9.2 | Sample Size Determination | 54 |
| 9.3 | Populations for Analyses | 54 |
| 9.4 | Statistical Analyses | 54 |
| 9.4.1 | General considerations. | 55 |
| 9.4.2 | Randomization and Stratification | 55 |
| 9.4.3 | Participant Disposition | 55 |
| 9.4.4 | Participant Demographics | 55 |
| 9.4.5 | Efficacy Analysis | 55 |
| 9.4.6 | Safety Analyses | 56 |
| 9.4.7 | Other Analyses | 56 |
| 9.5 | Interim Analysis | 57 |
| 9.6 | Data Safety Monitoring Board | 57 |
| 10. | SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS | 59 |
| 10.1 | Appendix 1 | 59 |
| 10.1.1 | Regulatory and Ethical Considerations | 59 |
| 10.1.2 | Financial Disclosure | 59 |
| 10.1.3 | Data Protection | 60 |
| 10.1.4 | Dissemination of Clinical Study Data | 60 |
| 10.1.5 | Source Documents | 61 |
| 10.1.6 | Study and Site Start and Closure | 61 |
| 10.1.7 | Publication Policy | 61 |
| 10.2 | Appendix 2 | 62 |
| 10.3 | Appendix 3 | 63 |
| 10.3.1 | Definition of Adverse Event and Adverse Reaction | 63 |
| 10.3.2 | Definition of Serious Adverse Event | 64 |
| 10.3.3 | Recording and Follow-Up of Adverse Event and/or Serious Adverse Event | 65 |
| 10.3.4 | Reporting of Serious Adverse Events | 66 |


| 10.4 | Appendix 4 | 67 |
|-----------|------------------------------------------------------------|----|
| 10.4.1 | Definitions | 67 |
| 10.4.2 | Contraception Guidance | 67 |
| 10.4.3 | Collection of Pregnancy Information | 68 |
| 10.5 | Appendix 5 | 70 |
| 11. | REFERENCES | 72 |
| | LIST OF TABLES | |
| Table 1: | Schedule of Assessments | 17 |
| Table 2: | Summary of Potential Risks Associated with VIS649 | 23 |
| Table 3: | Study Objectives and Endpoints | 28 |
| Table 4: | Study Interventions | 41 |
| Table 5: | Pharmacokinetic and Serum Immunoglobulin Sampling Schedule | 52 |
| Table 6: | Populations for Analysis | 54 |
| Table 7: | Scheduled Data Safety Monitoring Board Reviews | 57 |
| Table 8: | Protocol-Required Safety Laboratory Assessments | 62 |
| | LIST OF FIGURES | |
| Figure 1: | Study Design Schema | 16 |
| Figure 2: | Simulated Percent Baseline Immunoglobulin A by Dose | 35 |

# 1. PROTOCOL SUMMARY

# 1.1 Synopsis

| Name of Sponsor: Visterra, Inc. | | |
|---|---|---|
| Name of Investigational Intervention: VIS649 | | |
| Protocol Title: | A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Multiple Dose<br>Study to Evaluate the Efficacy and Safety of VIS649 in Participants with<br>Immunoglobulin A (IgA) Nephropathy (IgAN) | |
| Short Title: | Phase 2 Study of VIS649 for IgA Nephr | opathy |
| Rationale: | VIS649 is a humanized immunoglobulin G (IgG <sub>2</sub> ) monoclonal antibody that binds to and blocks the biological actions of the cytokine A PRoliferation Inducing Ligand (APRIL), a key factor in the production of aberrantly glycosylated IgA <sub>1</sub> (a-g- IgA <sub>1</sub> ), which is critical to the pathogenesis of IgAN. The central mechanism for the development of IgAN is the production of a-g IgA <sub>1</sub> . These a-g IgA <sub>1</sub> act as autoantigens and trigger formation of autoantibodies forming circulating immune complexes which deposit in the mesangium of the glomeruli and trigger an inflammatory response and complement activation, causing damage to the kidneys. In data from a single-ascending dose study of VIS649 in healthy volunteers, VIS649 reduced serum levels of IgA and a-g IgA <sub>1</sub> . The current study will test the hypothesis that blocking the biological actions of APRIL in IgAN patients leads to reduction of serum IgA (including a-g IgA <sub>1</sub> ) levels and will reduce or halt the progression of IgAN, as measured by decrease in proteinuria. The findings from this study will form the basis for subsequent clinical | |
| Objectives and | The key objectives and endpoints of the | study are: |
| Endpoints: | Primary Safety Objective | Primary Safety Endpoint |
| | To evaluate the safety and tolerability of multiple, monthly doses of VIS649 at each of 3 dosing levels, administered IV to IgAN participants over the course of 12 months as an add-on to SOC treatment with ACEI/ARB therapy, compared with saline placebo infusions as an add-on to SOC treatment with ACEI/ARB therapy | AEs graded by severity, clinical<br>laboratory tests, vital sign<br>measurements, and physical<br>examinations |

| <b>Primary Efficacy Objective</b> | Primary Efficacy Endpoint |
|---|---|
| To evaluate the dose response of multiple, monthly doses of VIS649 on proteinuria at each of 3 dosing levels, administered IV to IgAN participants over the course of 12 months as an add-on to SOC treatment with ACEI/ARB therapy, compared with saline placebo infusions as an add-on to SOC treatment with ACEI/ARB therapy | Change from baseline in uPCR (measured on natural log scale from 24-hour urine collection or the intended 24-hour urine collection) at Month 12 (ie, approximately 30 days after the twelfth dose is administered) |
| Secondary Objectives | Secondary Endpoints |
| <ul> <li>To evaluate the effect of repeated doses of VIS649 at 3 dosing levels versus placebo on the following parameters:</li> <li>uPCR at Month 9 and 15 (ie, 4 months following the final [12<sup>th</sup>] monthly dose administration)</li> </ul> | <ul> <li>Change from baseline in uPCR<br/>(measured on natural log scale<br/>from 24-hour urine collection or<br/>the intended 24-hour urine<br/>collection) at Months 9 and 15</li> </ul> |
| <ul> <li>24-hour urine protein excretion at Months 9, 12, and 15</li> <li>≥ 30% decline from baseline in uPCR at Months 9,12, and 15</li> <li>Clinical remission, defined as</li> </ul> | <ul> <li>Change from baseline in 24-hour urine protein excretion from baseline to Months 9, 12, and 15</li> <li>Participants in each group achieving a ≥ 30% decline from baseline in uPCR at Months 9, 12, and 15</li> </ul> |
| reduction in 24-hour urine protein excretion to < 300 mg/day for at least 3 consecutive months. | <ul> <li>Participants in each group<br/>achieving clinical remission</li> </ul> |
| • eGFR at Months 12 and 15 | • Change from baseline in eGFR at Months 12 and 15 |
| To evaluate the effect of repeated doses of VIS649 at each dosing level compared with placebo on the following PD parameters: IgA, IgG, and IgM concentrations | • Change from baseline in serum total IgA, IgG, and IgM concentrations at Months 9, 12, and 15 |
| To determine the PK profile of<br>repeated dose of VIS649, at each<br>dosing level | Serum PK parameters |
| To determine the PK/PD profile of<br>VIS649, relating VIS649 PK<br>parameters and biomarkers such as | Correlation of VIS649 PK parameters with changes in IgA, uPCR, and eGFR |

changes in IgA to changes in proteinuria and eGFR

• To screen for ADA responses

• Serum ADA levels

Abbreviations: ACEI = angiotensin-converting enzyme inhibitor; ADA = anti-drug antibody; AE = adverse event; a-g IgA = aberrantly glycosylated immunoglobulin A; APRIL= A PRoliferation Inducing Ligand; ARB = angiotensin receptor blocker; eGFR = estimated glomerular filtration rate; Ig = immunoglobulin; IgAN = immunoglobulin A nephropathy; IV = intravenous(ly); MEST = Mesangial cellularity, endocapillary proliferation, segmental sclerosis, tubular atrophy; PD = pharmacodynamic; PK = pharmacokinetic; SOC = standard of care; uACR = urinary albumin/creatinine ratio; uPCR = urinary protein/creatinine ratio.

#### Overall Design:

This is a Phase 2 multicenter, randomized, double-blind, placebo-controlled, multiple-dose study to evaluate the safety and efficacy of intravenously (IV) administered VIS649 over a 12-month treatment course in participants with IgAN. Participants will be enrolled from approximately 80 global sites in approximately 16 countries.

Screening evaluations, including physical examinations, vital signs, 12-lead electrocardiogram (ECG), safety laboratory testing (serum chemistry, hematology, urinalysis, serology, and pregnancy), and 24-hour urine collection, will take place approximately 30 days prior to the first dose of study intervention.

To be eligible, the participants should be on stable and maximally tolerated doses of either angiotensin-converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) therapy, as per standard of care (SOC) and applicable guidelines, for at least 3 months. Participants must be on at least 50% of the maximum recommended dose of the ACEIs or ARB to be considered as having adequate renin-angiotensin-aldosterone system (RAAS) blockade.

Participants who are unable to tolerate ACEI/ARB therapy may be eligible for participation in the study, if their overall management of IgAN, including blood pressure control, is as per SOC and applicable guidelines.

Enrolled participants must be adults, 18 years of age or older, with IgAN diagnosis confirmed by biopsy.

It is anticipated that most biopsies resulting in a diagnosis of IgAN will have been interpreted using the Mesangial cellularity, endocapillary proliferation, segmental sclerosis, tubular atrophy (MEST) (Cattran et al, 2009) or MEST-C scoring system (Trimarchi, Barratt et al. 2017) from the Oxford classification of IgAN.

A MEST-C score finding on kidney biopsy of T2 or C2 is exclusionary for this study. If the biopsy was not reported using the Oxford classification schema, the following findings are exclusionary: a) > 50% tubular atrophy, and/or b) > 25% crescents.

Participants must have Screening urinary protein/creatinine ratio (uPCR)  $\geq 0.75$  g/g or 24-hour urine protein  $\geq 1.0$  g/d, as measured from a 24-hour urine collection (or an intended 24-hour urine collection).

| | Participants must have estimated glomerular filtration rate (eGFR) |
|---|---|
| | ≥ 45 mL/min/1.73 m², calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula (Levey, Stevens et al. 2009). The study will evaluate 3 dose levels of VIS649 (2, 4, and 8 mg/kg) versus placebo. A total of 144 participants will be randomized with equal allocation (1:1:1:1) across the 4 intervention groups (approximately 36 participants per group). Randomization will be stratified first by region (Japan vs rest of world). |
| | A target of twelve or more participants are planned to be randomized in Japan; these participants will be randomized with equal allocation and without further stratification. The randomization for the rest of world will be stratified by screening uPCR ( $\leq 2.0 \text{ g/g vs} > 2.0 \text{ g/g}$ ). |
| | VIS649 or placebo will be administered as 12-monthly IV infusions starting on Day 1/Month 0. Participants will return to the study center on Day 8 and then monthly through Month 12 for safety, pharmacokinetic (PK) and/or pharmacodynamic (PD) assessments. |
| | Safety assessments will include review of adverse events (AEs) (including hypersensitivity reaction and anaphylactic reaction), physical examinations, injection site tolerability (including pain, irritation and tissue damage), clinical laboratory assessments (including biochemistry, hematology, and urinalysis), laboratory testing including serum Ig levels, vital sign measurements, and use of concomitant medications. |
| | Participants will return to the study center on Month 15, approximately 120 days following the last dose of study intervention (Dose 12) for additional safety, PK, PD, and efficacy assessments. Participants discontinuing dosing earlier will attend an early termination visit at the time of study intervention discontinuation and will be encouraged to attend the study visits as per schedule of assessments (SOA). |
| | It is anticipated that a roll-over extension study will be designed to enable longer term therapy for randomized participants. Further details will be provided in a separate protocol. |
| Number of Participants: | Approximately 144 participants. A target of twelve or more participants are planned to be randomized and enrolled in Japan. The remaining participants will be enrolled at sites in the rest of world; there are no country specific enrollment targets. |
| Intervention Groups and Duration: | The study will evaluate 3 dose levels of VIS649 (2, 4, and 8 mg/kg) versus placebo. VIS649 or placebo will be administered as a single, monthly IV infusion for 12 monthly doses. |
| | VIS649 will be administered IV over 1 hour, in a single, final volume 100 mL infusion in normal saline (0.9% NaCl), followed by a 25-mL saline flush. The dose of study intervention for the duration of the study will be based on the participant's Month 0 predose weight. |
| | Placebo (0.9% NaCl) will be administered IV over 1 hour as a single 100 mL infusion, followed by a 25 mL saline flush. |

An unblinded pharmacist will prepare drug or placebo for infusion. Participants, the Sponsor, the Investigator, and all other site study staff will be blinded to study intervention. The total study duration for each participant (from screening to end-of-study) will be up to 16 months [assuming 1 month for screening, 12 months for twelve monthly doses (including 30 days after the twelfth dose), and a 3-month safety follow-up]. **Target Population:** Key inclusion criteria for eligibility into the study are the following: 1. Participant is a male or female  $\geq$  18 years of age at the time of signing the informed consent. 2. Participants must have source verified biopsy-confirmed IgAN. 3. Participants has medical records showing that they have been on stable and maximally tolerated doses of either ACEI or ARB, as per SOC and applicable guidelines, for at least 3 months preceding screening. Participants should be on at least 50% of the maximum recommended dose of these agents to be considered as having adequate RAAS blockade. Participants who are unable to tolerate ACEI/ARB therapy may be eligible for participation in the study, if their overall management of IgAN, including blood pressure (BP) control, is as per SOC and applicable guidelines. 4. Participants must have screening uPCR  $\geq 0.75$  g/g measured from a 24-hour urine sample (or an intended 24-hour urine sample) or 24-hour urine protein  $\geq 1.0$  g/d, as measured from 24-hour urine sample (or an intended 24-hour urine sample). The proteinuria should be stable, defined as < 25% change when compared to values from  $\ge 3$  months previously (if available). If previous values are not available or if the change from a prior value is > 25%, a repeat measurement of proteinuria will be done after 15 days and the participant should fulfill the above proteinuria criteria to be eligible for randomization in the study. The proteinuria should be assessed when the participant is considered to be in steady state with no recent heavy exercise, fever, or other potential issues that could impact the result. 5. Participants must have eGFR  $\geq$  45 mL/min/1.73 m<sup>2</sup>, calculated using the CKD-EPI formula. The eGFR should be stable, as defined by a < 25% change when compared to values from  $\ge 3$  months previously (if available). If previous values are not available or if the change from a prior value is > 25%, a repeat measurement of eGFR will be done after 15 days and the participant should fulfill the eGFR criteria to be eligible for randomization in the study. The eGFR should be measured when the participant is considered to be in a steady state without recent changes in volume status, medications that could impact the result (eg, nonsteroidal anti-inflammatory drugs [NSAIDs], aminoglycosides, co-trimoxazole) or changes in dietary protein intake.

6. Participant's serum Ig values must meet the criteria below:

a.  $IgG: \ge 700 \text{ mg/dL}$ b.  $IgM: \ge 40 \text{ mg/dL}$ 

c.  $IgA: \ge 70 \text{ mg/dL}$ 

#### Key exclusion criteria:

- 1. Participant has secondary forms of IgAN as defined by the treating physician (eg, Henoch-Schönlein purpura, minimal change disease with IgA deposits, infections associated with IgAN or IgAN associated with hepatic cirrhosis).
- 2. Participant has co-existing chronic kidney disease, other than IgAN.
- 3. Participant has evidence of additional pathological findings in the kidney biopsy (eg, diabetic kidney disease, membranous nephropathy, or lupus nephritis lupus). However, hypertensive vascular changes are acceptable.
- 4. Participant has kidney biopsy MEST or MEST-C score of T2 or C2 from the Oxford IgAN classification schema. If MEST-scoring was not performed, the presence of > 50% tubulointerstitial fibrosis, or crescents in > 25% of glomeruli is exclusionary.
- 5. Participant has nephrotic syndrome, defined for this purpose as 24-hour urine protein > 3.5 g with concurrent hypoalbuminemia (serum albumin < 2.5 g/dL), hyperlipidemia (total cholesterol > 350 mg/dL), and edema.
- 6. Participant has received a solid organ transplant, including kidney.
- 7. Participant has received bone marrow or hematologic stem cell transplantation
- 8. Participant is currently receiving systemic immunosuppression (excluding topical, ophthalmic, per rectum or inhaled corticosteroids).
- 9. Participant has received systemic steroids within the 12 weeks prior to initial screening.
- 10. Participant has received treatment with 2 or more systemic immunosuppressive agents within 2 years prior to initial screening
- 11. Participant has chronic infectious diseases (eg, chronic urinary tract infection, chronic sinusitis, bronchiectasis, active pulmonary or systemic tuberculosis, chronic viral hepatitis, hepatitis C virus or hepatitis B virus or HIV infection).
- 12. Participant has acute infectious disease at the time of screening.

  Participants may be rescreened following resolution of acute infection (such as urinary tract infection or respiratory tract infection), provided there is no evidence of an immunosuppressive condition that predisposed the participant to this infection.
- 13. Participant has Type 1 diabetes.

| | 11 - 1 - | |
|---|---|---|
| | 14. Patient has uncontrolled Type 2 diabetes, as evidenced by a screening hemoglobin A1c value > 8%. | |
| | 15. Participant has uncontrolled blood pressure (> 160 mm Hg systolic or > 110 mm Hg diastolic) | |
| | 16. Participant has a history of chronic autoimmune neurodegenerative disorders such as multiple sclerosis. | |
| Data Safety<br>Monitoring Board: | An independent data safety monitoring board (DSMB) will review unblinded safety data. The DSMB will meet at 5 scheduled data review meetings and on an ad hoc basis as needed. Details regarding the content and scope of safety assessments, as well as the governing of the DSMB, will be described in a separate DSMB charter. | |
| | Data safety monitoring boar requirements are met: | ard meetings will be scheduled as the following |
| | Scheduled DSMB Review | Number of Participants and Treatment Exposure |
| | DSMB review #1 | Scheduled once 12 participants have been randomized and have completed at least 3 months of dosing. |
| | DSMB review #2 Scheduled once 24 participants have been randon and have completed at least 3 months of dosing. DSMB review #3 Scheduled once ~25% of participants have been randomized and have completed 3 months of dos | |
| | DSMB review #4 Scheduled once ~50% of participants have been randomized and have completed 6 months of dosing and ~ 20 participants have completed 12 months of dosing | |
| | DSMB review #5 | Scheduled once ~50% of participants have been randomized and have completed 12 months of dosing. |
| | Abbreviations: DSMB = dat | a safety monitoring board. |
| Statistical Methods: | General Considerations | |
| | All data collected will be documented using summary tables, figures, and/or data listings presented by intervention and dose group. For continuous variables, descriptive statistics (number [n], mean, geometric mean and coefficient of variation [%CV], as appropriate, median, standard deviation, minimum, and maximum) will be presented. For categorical variables, frequencies and percentages will be presented. As appropriate, a 95% CI will be presented. Graphical displays may be presented. | |
| | Randomization and Stratifi | cation |
| | ally assigned in a 1:1:1:1 ratio to receive VIS649 at 2, with approximately 36 participants randomized per mization will be stratified first by region (Japan vs rticipants will be randomized with equal allocation cation. Randomization for the rest of world will then | |

be stratified by screening uPCR ( $\leq 2.0 \text{ g/g vs} > 2.0 \text{ g/g}$ ).

Interim Analysis

In addition to 5 DSMB safety reviews, 3 interim PK/Ig analyses and 1 interim efficacy analysis are planned. The interim PK/Ig analyses will provide additional data for population PK/PD modeling and will advise the study Sponsor on future study design and planning.

An interim efficacy analysis will be performed at the time of the fourth scheduled DSMB meeting (when 50% of randomized participants have completed the Month 6 visit reflecting 6 months of study intervention or placebo exposure and  $\sim 20$  participants have completed 12 months of dosing). Group-unblinded efficacy summaries (with individual participant treatment blinded) will be prepared for Sponsor review to inform future study design.

The interim efficacy analysis will not include hypothesis testing and will be for the purpose of future study design and planning. The primary efficacy endpoint, change in proteinuria from baseline, will be analyzed. No modifications to this study protocol are planned based on results of the interim analyses.

#### Planned analyses

The primary efficacy outcome for this study is the change from baseline in uPCR on the natural log scale at Month 12. Dose response will be explored using orthogonal contrasts. Sensitivity analysis will follow using dose as a continuous covariate with associated linear, quadratic, and cubic terms.

In addition, to assess the dose response over time, a Mixed Model with Repeated Measurements (MMRM) which includes fixed class-effects of treatment, visit, randomization strata, and treatment by visit interaction, with a fixed effect covariate of baseline uPCR on the natural log scale will be used. An unstructured variance covariance matrix will be assumed, and linear, quadratic, and cubic dose responses will be assessed.

Secondary efficacy endpoints will be summarized using descriptive statistics. In addition, comparisons between dose groups against placebo will be performed using Analysis of Covariance or MMRM for continuous measures and logistic regression or generalized estimating equations for categorical variables.

Safety will be assessed by evaluation of AEs (including hypersensitivity reaction and anaphylactic reaction), physical examinations, injection site tolerability (including pain, irritation and tissue damage), clinical laboratory assessments (including biochemistry, hematology, and urinalysis), laboratory testing including serum Ig levels, vital signs, and concomitant medications.

Analysis of PK parameters will include participant data-listings of serum concentrations and summary statistics by group including means, geometric means, standard deviations, %CV, medians, and ranges, as appropriate. Summary graphs including mean concentration-time profiles by group will also be presented. For the subset of participants for whom intensive PK samples are collected, serum concentration data will be analyzed by

. In addition,

| as implemented in NONMEM or equivalent software. Additional |
|-------------------------------------------------------------|
| analyses and summaries may be generated as appropriate. |

#### 1.2 Schema

Figure 1: Study Design Schema



Abbreviations: ACEI = angiotensin-converting enzyme inhibitor; ARB = angiotensin receptor blocker; eGFR = estimated glomerular filtration rate; uPCR = urine protein to creatinine ratio.

CONFIDENTIAL VIS649-201 Protocol Version 0.2

# 1.3 Schedule of Assessments

**Table 1:** Schedule of Assessments

| Procedures | Scr1 | Intervention Period (Study Month) EO | | | | | | | | | | | | EOS <sup>2</sup> | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Month | N/A | | M0 | | | | М3 | M4 | M5 | M6 | M7 | M8 | М9 | M10 | M11 | M12/<br>ET <sup>3</sup> | M15 |
| Nominal Study Day | -301 | D1 Pre infusion | D1 Post infusion | D8 | D30 | D60 | D90 | D120 | D150 | D180 | D210 | D240 | D270 | D300 | D330 | D360 | D450 |
| Visit allowance (±days) | | N/A | N/A | ±3 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 |
| Study Visit | N/A | 1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 |
| Informed consent | X | | | | | | | | | | | | | | | | |
| Inclusion/exclusion criteria review | X | X | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | | |
| Review of kidney biopsy <sup>4</sup> | X | | | | | | | | | | | | | | | | |
| Physical examination <sup>5</sup> | X | | | | | | | | | | | | | | | X | |
| Weight | X | X | | | | | | | | X | | | X | | | X | X |
| Vital signs <sup>6</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| 12-lead ECG | X | | | | | | | | | | | | | | | | |
| Randomization | | X | | | | | | | | | | | | | | | |
| Study intervention infusion <sup>7</sup> | | 2 | K | | Х | х | х | х | х | X | X | х | X | Х | х | | |
| AE monitoring | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | Х | X |
| Concomitant medications review | Х | х | х | X | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х | Х |
| HBV, HCV, HIV<br>serology | Х | | | | | | | | | | | | | | | | |
| Serum β-hCG (females only) | Х | | | | | | | | | | | | | | | | |
| Urine β-hCG (females only) | | х | | | Х | Х | Х | Х | Х | Х | х | Х | Х | Х | Х | Х | Х |
| Serum chemistry <sup>8</sup> | Х | Х | | | Х | х | х | х | Х | Х | Х | х | х | Х | Х | Х | Х |
| Hematology <sup>9</sup> | X | х | | | | | X | | | Х | | | | X | | х | Х |

| Procedures | Scr1 | rl Intervention Period (Study Month) | | | | | | | | | | | EOS <sup>2</sup> | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Month | N/A | | M0 | | M1 | M2 | М3 | M4 | M5 | M6 | M7 | M8 | M9 | M10 | M11 | M12/<br>ET <sup>3</sup> | M15 |
| Nominal Study Day | -301 | D1 Pre infusion | D1 Post infusion | D8 | D30 | D60 | D90 | D120 | D150 | D180 | D210 | D240 | D270 | D300 | D330 | D360 | D450 |
| Visit allowance (±days) | | N/A | N/A | ±3 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 |
| Study Visit | N/A | 1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 |
| Urinalysis (dipstick and microscopy) <sup>10</sup> | X | Х | | X | Х | Х | Х | Х | Х | Х | X | Х | Х | Х | Х | Х | х |
| 24-hour urine collection <sup>11</sup> | X | | | | | | | | | | | | X | | | Х | х |
| Urine sample for uPCR determination | x <sup>12</sup> | Х | | X | Х | Х | X | X | Х | Х | X | Х | x <sup>12</sup> | Х | X | x <sup>12</sup> | x <sup>12</sup> |
| Urine sample for uACR determination | x <sup>12</sup> | | | | | | | | | | | | x <sup>12</sup> | | | x <sup>12</sup> | x <sup>12</sup> |
| Blood sample for lymphocytes | | х | | | | | | | | Х | | | | | | X | х |
| Serum for PK <sup>13</sup> | | X | х | х | x <sup>14</sup> | x <sup>14</sup> | x <sup>14</sup> | x <sup>14</sup> | x <sup>14</sup> | x <sup>14</sup> | x <sup>14</sup> | x <sup>14</sup> | x <sup>14</sup> | x <sup>14</sup> | x <sup>14</sup> | х | х |
| Blood for total IgA, IgG, and IgM <sup>13</sup> | х | х | х | X | Х | х | х | х | х | х | | х | х | х | х | х | х |
| Blood for IgA subtypes | | X | | | | | Х | | | Х | | | Х | | | Х | х |
| Serum for APRIL <sup>1</sup> | | X | х | | X | Х | x <sup>14</sup> | Х | Х | x <sup>14</sup> | Х | X | x <sup>14</sup> | х | x <sup>14</sup> | Х | х |
| Serum for a-g IgA <sub>1</sub> and anti-IgA <sub>1</sub> | Х | Х | | | | | х | | | Х | | | Х | | | Х | х |
| Serum for ADA <sup>15</sup> | | X | | | X | Х | | Х | | Х | | Х | | | Х | Х | х |
| Blood sample for DNA <sup>16</sup> | | X | | | | | | | | | | | | | | | |
| Urine sample for exploratory biomarker assessments <sup>17</sup> | | Х | | | | | Х | | | Х | | | Х | | | х | х |
| Blood for markers of complement activity <sup>13</sup> | | х | | | | | | | | Х | | | | | | х | |
| Saliva samples for IgA levels | | х | | | | | | | | Х | | | | | | х | |

Abbreviations: ACEI = angiotensin-converting enzyme inhibitor; ADA = anti-drug antibody; AE = adverse event; a-g IgA = aberrantly glycosylated immunoglobulin A; APRIL= A PRoliferation Inducing Ligand; ARB = angiotensin receptor blocker; β-hCG = beta-human chorionic gonadotropin; BAFF = B-cell activating factor; BP = blood

pressure; D = Day; ECG = electrocardiogram; eCRF = electronic case report form; EOS = end-of-study; ET = early termination; HBV = hepatitis B virus; HCV = hepatitis C virus; HIV = human immunodeficiency virus; HR = heart rate; Ig = immunoglobulin; IgAN = immunoglobulin A nephropathy; M = Month; N/A = not applicable; PD = pharmacodynamics; PK = pharmacokinetics; RR = respiratory rate; Scr = screening; SOC = standard of care; uACR = urinary albumin/creatinine ratio; uPCR = urinary protein/creatinine ratio.

- All participants will undergo screening. To be eligible, participants should be on stable and maximally tolerated treatment with either ACEI or ARB, as per SOC and applicable guidelines, for at least 3 months. Participants who are unable to tolerate ACEI/ARB therapy may be eligible for participation in the study, if their overall management of IgAN, including BP control, is as per SOC and applicable guidelines.
- Participants must complete EOS assessments approximately 120 days after the last dose of study intervention. Participants discontinuing early will be encouraged to attend study visits as per the schedule, including the EOS visit. Adverse event and concomitant medication monitoring should be performed through the EOS visit; AEs that are ongoing at EOS should be monitored until resolution or 30 days after the EOS, whichever is shorter.
- Participants discontinuing early must complete ET assessments at the time of treatment discontinuation.
- 4 A biopsy diagnostic of IgAN must have been performed and source-verified documentation must be available.
- A complete physical examination, to include assessments of the cardiovascular, respiratory, gastrointestinal and neurological systems will be completed at the screening and end-of-treatment visit.
- Witals signs include BP, HR, RR, and temperature. Vital signs measurements on dosing days will be recorded within 15 (±5) minutes prior to the start of the infusion, every 15 minutes until the infusion is complete, and 60 minutes and 2 hours postinfusion.
- The dose of study intervention will be based on the M0 predose weight.
- The comprehensive list of serum chemistry tests to be performed is provided in Appendix 2. A full serum chemistry panel will be obtained at screening and on M0, M3, M6, M9, M12, and M15; the following tests are required at other visits: sodium, potassium, chloride, bicarbonate, blood urea nitrogen, creatinine, and glucose. Local laboratory assessments may be performed at Investigator discretion throughout the study in the course of patient care (but not assessments that would potentially unblind treatment status, such as measurement of immunoglobulin levels). Any clinically significant abnormalities should be recorded in the eCRF.
- The comprehensive list of hematology tests to be performed is provided in Appendix 2.
- The comprehensive list of urinalysis tests to be performed is provided in Appendix 2. On days of 24-hour urine collection, the uPCR sample will be collected from the 24-hour urine collection and routine urinalysis will be performed on a sample freshly voided during the clinic visit.
- Participants will discard the first void and begin a 24-hour urine collection the day prior to the clinic visit. For all 24-hour urine collection, the following parameters will be obtained or derived: 24-hour urine volume, protein, albumin, and creatinine, uPCR, and uACR.
- Samples should be taken from the 24-hour urine sample.
- Up to 60 participants (approximately 15 per cohort) may have a more extensive PK and PD sampling schedule, as described in Table 5. Study participants agreeing to participate in this more intensive PK and PD sample collection sub-study will sign an additional informed consent for this activity.
- Blood samples to be collected before and after study intervention infusion at all visits.
- Samples for ADA assessment will be collected before the start of infusion.
- 6 Samples for evaluation of host genetic markers related to IgAN susceptibility loci, the APRIL/BAFF pathway, and/or immunity will be collected before the start of infusion.
- On days of 24-hour urine collection, urine samples for exploratory biomarker analysis will be collected and stored from a sample freshly voided during the clinic visit.

#### 2. INTRODUCTION

VIS649 is a humanized IgG<sub>2</sub> monoclonal antibody being developed for the treatment of immunoglobulin A nephropathy (IgAN), an autoimmune glomerulonephritis characterized by the deposition of immunoglobulin A (IgA)-containing immune complexes in the kidney.

#### 2.1 Study Rationale

Immunoglobulin A nephropathy is a chronic disease affecting the kidneys. It is clinically characterized by proteinuria, hematuria and progressive decline of glomerular filtration rate (GFR). IgAN is characterized histologically by dominant or co-dominant deposition of IgA in the kidney glomerulus (Rodrigues, Haas et al. 2017). The central mechanism for the development of IgAN is the production of aberrantly glycosylated IgA<sub>1</sub> (a-g IgA<sub>1</sub>) which has been attributed to a combination of genetic and environmental factors. These a-g IgA<sub>1</sub> act as auto-antigens and trigger formation of autoantibodies forming circulating immune complexes which deposit in the mesangium of glomeruli and trigger an inflammatory response and complement activation (Kiryluk, Moldoveanu et al. 2011, Berthoux, Suzuki et al. 2012, Kiryluk, Novak et al. 2013, Kiryluk, Li et al. 2014, Kiryluk and Novak 2014). This results in episodic and cumulative kidney damage. Natural history studies indicate that IgAN may progress to end stage kidney disease in approximately 30% of patients, over the course of 10 years (Lai, Tang et al. 2016).

Proteinuria is an important marker of progression of renal disease in patients with IgAN. Patients with significant proteinuria (> 1.0 g/day) have a faster decline of eGFR and progression to end-stage renal disease (ESRD), when compared to patients with lower degrees of proteinuria (< 500 mg/day). Hence reduction in proteinuria is a crucial aspect in the management of IgAN (Reich, Troyanov et al. 2007, Nam, Kie et al. 2014, Inker, Mondal et al. 2016).

The cytokine A PRoliferation Inducing Ligand (APRIL), which belongs to the tumor necrosis factor ligand superfamily, has emerged as a key factor in the pathogenesis of IgAN through mediation of the immunoglobulin isotype switch during B-cell development, production of IgA, plasma-cell survival, and possibly specifically influencing production of a-g IgA<sub>1</sub> as well (Castigli, Scott et al. 2004, Varfolomeev, Kischkel et al. 2004, Endo, Nishio et al. 2007, Bossen, Cachero et al. 2008). Studies in IgAN patients have shown that elevated APRIL levels correlate with poor kidney outcomes, when compared with patients with lower APRIL levels (Han, Yang et al. 2016, Zhai, Zhu et al. 2016). A similar trend is also seen with a-g IgA<sub>1</sub> levels, with higher levels associated with faster and more frequent progression to kidney failure when compared to patients with lower a-g IgA<sub>1</sub> levels (Castigli, Scott et al. 2004, Berthoux, Suzuki et al. 2012, Zhao, Hou et al. 2012).

VIS649 is a humanized IgG<sub>2</sub> monoclonal antibody (mAb) that binds to and blocks the biological actions of APRIL, preventing its binding to its receptors, transmembrane activator and CAML interactor (TACI), and B-cell maturation antigen (BCMA). Blocking the biological actions of APRIL reduces the production of IgA. The hypothesis to be tested in this study is that a decrease in the production of IgA and a-g IgA<sub>1</sub> will diminish the formation of circulating immune complexes and their deposition in the glomeruli, allowing injury repair and clinical improvement, as measured by reduction in proteinuria.

In data from a single-ascending dose study (VIS649-101) of VIS649 in healthy participants, VIS649 reduced serum levels of IgA and a-g IgA<sub>1</sub>. The current study will test the hypothesis that blocking the biological actions of APRIL in IgAN patients leads to reduction of serum IgA (including a-g IgA<sub>1</sub>) levels and will reduce or halt the progression of IgAN as measured by reduction in proteinuria (the study's primary efficacy endpoint). The current study will also assess the safety of VIS649 in patients with IgAN and collect extensive data on pharmacokinetics (PK) and pharmacodynamics (PD).

The findings from this study will form the basis for subsequent clinical development of VIS649.

#### 2.2 Background

Immunoglobulin A nephropathy is one of the most common primary glomerular diseases and affects patients globally, with some geographical variation in incidence and prevalence (Wyatt and Julian 2013, Rodrigues, Haas et al. 2017, Schena and Nistor 2018). Clinical presentation varies from incidentally detected asymptomatic hematuria and proteinuria to rapidly progressive glomerulonephritis requiring dialysis. Immunoglobulin A nephropathy is a significant cause of chronic kidney disease (CKD) and ESRD, with 30–40% of patients reaching ESRD 20–30 years after the first clinical presentation. Immunoglobulin A nephropathy can occur in either sporadic (90–95%) or familial (5%–10%) patterns. Patients with familial IgAN might have poorer prognoses than those with sporadic disease, with an increased risk of progression to renal failure (Lai, Tang et al. 2016).

Immunoglobulin A nephropathy is diagnosed by kidney biopsy, which shows dominant or co-dominant IgA deposition on immunofluorescence. The pathogenesis of IgAN is currently thought to be a multi-hit process, the "first hit" being the production of a-g-IgA<sub>1</sub>. The primary defect is the deficiency of galactose in the hinge region of IgA<sub>1</sub>. As a consequence, the N-acetylgalactosamine in the truncated IgA<sub>1</sub> hinge region glycan is exposed and acts as an autoantigen. Multiple cohort studies have shown the relationship between elevated a-g IgA<sub>1</sub> and IgAN, with higher a-g IgA<sub>1</sub> levels having more rapid disease progression. The "second hit" consists of IgA and IgG auto-antibody production against these a-g IgA<sub>1</sub>. The "third hit" consists of formation of circulating immune complexes consisting of the IgG/IgA auto antibody and a-g IgA<sub>1</sub> antigen complex. The "fourth hit" consists of deposition of these circulating immune complexes in the mesangium of the glomeruli. These antigen-antibody complexes are nephritogenic and trigger an inflammatory response leading to infiltration of macrophages, monocytes and T cells, local release of cytokines, complement activation and activation of renin-angiotensin cascade. This leads to glomerular injury and tubulointerstitial fibrosis, clinically manifesting as proteinuria, hematuria, hypertension and reduced GFR (Berthoux, Suzuki et al. 2012, Floege, Moura et al. 2014, Knoppova, Reily et al. 2016, Mestecky, Novak et al. 2016).

Proteinuria is a common manifestation of IgAN and the degree of proteinuria correlates with disease progression, with faster decline of estimated glomerular filtration rate (eGFR) and progression to ESRD in patients with high-grade proteinuria (> 1.0 gm/day) when compared to patients with low-grade proteinuria (< 0.5 gm/day) (Reich, Troyanov et al. 2007, Nam, Kie et al. 2014, Inker, Mondal et al. 2016, Thompson, Carroll et al. 2019). Control of proteinuria is a key therapeutic target in patients with IgAN. Measures to control proteinuria often consist of renin-angiotensin-aldosterone system (RAAS) blockade in the form of angiotensin-converting

enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) therapy, blood pressure (BP) control, statins to control cholesterol, smoking cessation, low-salt diet, low-protein diet and avoidance of nephrotoxic drugs. If patients continue to have significant proteinuria despite these measures, they are usually treated with nonspecific immunosuppressive agents such as steroids, azathioprine, mycophenolate mofetil, or cyclophosphamide (Boyd, Cheung et al. 2012, KDIGO 2012, Radhakrishnan and Cattran 2012, Barbour and Feehally 2017, Rodrigues, Haas et al. 2017). These drugs, especially steroids (Pozzi, Andrulli et al. 2004, Rauen, Eitner et al. 2015, Tesar, Troyanov et al. 2015, Lv, Zhang et al. 2017) have been shown to be beneficial from a renal perspective in some studies, but their use is often complicated by significant adverse effects such as increased risk of infections, metabolic derangements, cosmetic changes, weight gain, fractures, and neuropsychiatric manifestations. Some of these agents have other significant risks such as increased risk of malignancies with prolonged administration. The significant side effects of these drugs preclude chronic use of these agents and limit their benefits in a chronic disease such as IgAN.

APRIL is a member of the tumor necrosis factor (TNF) superfamily of ligands and is emerging as a key mediator in IgAN pathogenesis and disease progression based on a convergence of genetic, biochemical, and clinical data. APRIL is produced by myeloid and mucosal epithelial cells. APRIL regulates B cell-mediated immune responses through several mechanisms, including class-switch recombination, principally through its 2 receptors, TACI and BCMA. APRIL is also important for plasmablast differentiation in secondary lymphoid organs. In addition, myeloid-derived APRIL mediates plasma cell survival by promoting the formation of so-called "survival niches" within the bone marrow microenvironment and mucosal compartments, leading to the establishment of a reservoir for long-lived antibody-secreting cells (Bossen, Cachero et al. 2008).

Evidence of the critical role of APRIL in IgAN includes the following: (a) serum a-g IgA<sub>1</sub> (auto-antigen) levels are elevated in patients with IgAN and correlate with APRIL levels and disease severity; (b) genome-wide association studies link APRIL to the disease; (c) serum APRIL is elevated in patients with IgAN and higher APRIL levels among IgAN patients are associated with more rapid progression to kidney failure (Mestecky, Raska et al. 2013, Han, Yang et al. 2016, Muto, Manfroi et al. 2017).

In a mouse model of IgAN, administration of an anti-APRIL antibody similar to VIS649 led to lower IgA deposits in the kidney, lower proteinuria, and less glomerular sclerosis compared with animals administered a control antibody that does not bind APRIL. These data suggest that APRIL plays a key role in the pathogenesis of IgAN and that blocking APRIL could be an attractive approach for the treatment of IgAN (Myette, Kano et al. 2019).

VIS649 is a humanized IgG<sub>2</sub> mAb against the biologically active form of APRIL. VIS649 was tested in healthy human participants in a Phase 1, randomized, placebo-controlled, single-ascending dose first-in-human study to assess the safety, tolerability, PK and PD of VIS649 (Study VIS649-101). The study enrolled 51 participants in 5 sequential dosing cohorts. Participants in Cohorts 1 to 4 received 4 different dose levels of VIS649 (0.5, 2.0, 6.0, and 12 mg/kg respectively), enrolling 9 participants per cohort (7 participants receiving VIS649 and 2 participants receiving placebo). Cohort 5 had 15 participants with 10 receiving VIS649 and 5 participants receiving placebo. Participants in Cohort 5 received 6.0 mg/kg of VIS649 on Day 1 and subsequently received a tetanus and diphtheria (Td) vaccine on Day 28. Blinded group

data are available, including IgA levels. Preliminary data show that the total serum IgA declined by up to 70% from normalized baseline values in these healthy participants. The vaccine response in Cohort 5 was intact, with a comparable IgG response to Td vaccine in participants receiving VIS649 and participants receiving placebo. Mean serum IgG levels declined by up to 30% below normalized baseline values and mean immunoglobulin M (IgM) levels showed a marked decline and were up to 80% below the normalized levels. These declines in the immunoglobulin (Ig) levels were reversible and the time taken to restoration of the Ig levels to baseline was dependent on the dose of VIS649, with higher doses requiring a longer time period. VIS649 was very well tolerated across all dose levels and there were no serious adverse events (SAEs) attributed to VIS649. Further details can be found in the Investigator's Brochure.

The adverse risk—benefit ratio of nonspecific immunosuppressive agents, preclude the chronic use of such agents and highlight the need for the development of an effective alternative that acts specifically at relevant pathophysiological factors in IgAN and is also likely safe for chronic use.

#### 2.3 Benefit/Risk Assessment

#### 2.3.1 Risk Assessment

Table 2 summarizes the important potential risks that have been recognized during the conduct of VIS649 nonclinical and clinical development programs. At present, all are considered potential risks.

More detailed information about the risks and reasonably expected adverse events (AEs) of VIS649 may be found in the Investigator's Brochure.

Table 2: Summary of Potential Risks Associated with VIS649

| Potential Risk of<br>Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| IgA suppression risk | Based on the mechanism of action of VIS649, preclinical studies, and human data from healthy volunteers, total serum IgA levels are expected to be suppressed to nadir levels There is increasing recognition that selective IgA deficiency, which has typically been associated with IgA levels below the lower limit of detection may be associated with recurrent sinopulmonary infection, allergy, autoimmunity, and gastrointestinal microbiome perturbation (Yazdani, Azizi et al. 2017, Fadlallah, El Kafsi et al. 2018). VIS649 is expected to reduce but not ablate IgA expression. Additionally, the syndrome of selective IgA deficiency is often associated with additional immunologic impairments, including T-cell disorders which are not expected to occur with VIS649 dosing. | Serum IgA, IgG, and IgM will be measured on a monthly basis (as blinded data, to be made available for routine DSMB review). The DSMB will assess unblinded safety data on a scheduled and ad hoc basis as needed, including AEs, laboratory data and Ig data. The DSMB charter calls for assessment of the relationship of AEs to observed Ig levels (IgA, IgG and IgM) in study participants. If needed, the DSMB charter also calls for specific risk-mitigation strategies including, but not limited to, change in inclusion/exclusion criteria, establishing criteria for stopping study intervention in a participant or a cohort, |

| D-442-1 D/-16 | 1 | 1 |
|---|---|---|
| Potential Risk of<br>Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
| | Additional information can be found in the Investigator's Brochure. | establishing criteria for rescue<br>therapies such as IVIG and<br>change in dosing schedule of a<br>participant or a cohort based<br>on standardized safety lab<br>analysis and AE analysis. |
| IgG suppression risk | VIS649 is expected to have a moderate effect on serum IgG levels In the most commonly occurring disease state characterized by hypogammaglobulinemia, CVID, total IgG levels at diagnosis are typically below 250 mg/dL. CVID has been associated with recurrent otitis media, chronic sinusitis, and recurrent pneumonia, which may result in bronchiectasis (Ballow 2002, Furst 2009). The risk of these complications with VIS649 therapy is considered low, given the multifaceted immunologic dysfunction associated with CVID in comparison with the moderate (but not profound) anticipated effect of VIS649 on serum IgG. Additional information can be found in the Investigator's Brochure. | <ul> <li>Please see above regarding Ig and AE data monitoring under DSMB review.</li> <li>To further reduce the risk of persistent clinically impactful suppression of IgG, the protocol inclusion criteria require an IgG level &gt; 700 mg/dL at screening for enrollment</li> <li>In a Phase 1 study of VIS649 in healthy participants, IgG responses to recall challenge with tetanus and diphtheria toxoid vaccination was comparable between recipients receiving placebo and VIS649.</li> <li>In preclinical toxicology studies performed in nonhuman primates, the ability to generate a de novo humoral immune response to a novel T-cell dependent antigen (keyhole limpet hemocyanin) was not suppressed by VIS649, and peripheral blood myeloid cell line populations were unaffected.</li> </ul> |
| IgM suppression risk | Based on the mechanism of action of VIS649, preclinical studies, and human data from healthy volunteers, total serum IgM is expected to be suppressed to levels approximately below baseline. Most patients with selective IgM deficiency are asymptomatic, but a few patients develop chronic and recurrent infections and | Please see above regarding Ig and AE data monitoring under DSMB review. |

| Potential Risk of<br>Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| | increased risk of auto-immune diseases(Yel, Ramanuja et al. 2009, Louis and Gupta 2014, Louis, Agrawal et al. 2016, Janssen, Macken et al. 2018). Selective IgM deficiency is usually associated with other defects such as decreased T-helper cell activity, increased isotype specific suppressor T cells, increased CD8 Treg cells, and intrinsic B cell defects. VIS649 is not expected to have effects such as these on cellular immunity. | |
| Nonspecific immunosuppression risk | There is the possibility of nonspecific immunodeficiency with potential risk of exacerbation of pre-existing latent infection or poor response to new infection. Additional information can be found in the Investigator's Brochure. | <ul> <li>Participants with acute or chronic infections at the time of screening are prohibited from enrollment.</li> <li>Participants with underlying iatrogenic or primary immunodeficiency syndromes are prohibited from enrollment.</li> <li>DSMB monitoring will include careful attention to infection-related AEs.</li> <li>Concurrent treatment with systemic corticosteroids or other immunosuppressive therapy is prohibited during study conduct.</li> </ul> |
| Infusion reactions (anaphylaxis, fever, chills, rigors, nausea, vomiting, pain, headache, dizziness, shortness of breath, bronchospasm, hypotension, hypertension, pruritus, rash, urticaria, angioedema, diarrhea, tachycardia, and chest pain) | There was no effect of VIS649 on measured plasma cytokine concentrations in the monkey toxicology studies, and VIS649 did not stimulate significant cytokine release in an in vitro human peripheral blood lymphocyte cytokine release assay. There were no SAEs attributable to VIS649 among participants in the Phase 1 VIS649-101 study at dose levels up to 12 mg/kg. Severe infusion reactions such as anaphylaxis have not been observed with VIS649 in humans. Additional information can be found in the Investigator's Brochure. | All VIS649 doses will be administered at the clinical site by trained personnel, and participants will be closely monitored for the occurrence of infusion reactions. |
| Delayed allergic reactions<br>(SSLR [ie, urticaria,<br>fever, general glandular<br>enlargement, joint pains]) | Delayed allergic reactions to a mAb such as serum sickness (ie, urticaria, fever, general glandular enlargement, joint pains) have been reported with other mAb's and may not appear until several days or weeks after the infusion. Additional information can be found in the Investigator's Brochure. | Participants will be monitored for AEs throughout the duration of the study. |

| Potential Risk of<br>Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Injection site reactions | Injection site reactions may occur following administration of any intravenous therapy. | All VIS649 doses will be administered at the clinical site by trained personnel, and participants will be closely monitored for injection site reactions. |

Abbreviations: AE = adverse event; APRIL= A Proliferation Inducing Ligand; CVID = common variable immunodeficiency; DSMB = data safety monitoring board; Ig = immunoglobulin; IgA = immunoglobulin A; IgG = immunoglobulin G; IgM = immunoglobulin M; IVIG = intravenous immunoglobulin; LLN = lower limit of normal; mAb = monoclonal antibody; PD = pharmacodynamic(s); PK = pharmacokinetic(s); SAE = serious adverse event; SSLR = serum-sickness like reaction.

#### 2.3.2 Benefit Assessment

Immunoglobulin A nephropathy is a chronic disease with periodic flares. IgAN is a significant cause of chronic kidney disease (CKD) and ESRD, the clinical progression varies, with 30 – 40% of patients reaching ESRD 20 to 30 years after the first clinical presentation (Lai, Tang et al. 2016). These patients have significantly increased mortality and morbidity, with life expectancy reduced by 6 to 10 years when compared to healthy individuals. (Hastings, Bursac et al. 2017, Jarrick, Lundberg et al. 2019). There are currently no approved therapies for IgAN, and the current treatment strategies consist of 2 main aspects: nonspecific supportive treatments consisting of blood pressure control, treatment with ACEI/ARB, smoking cessation, lipid reduction, low-salt diet, or fish oil and immunosuppressive therapies such as steroids, cyclophosphamide, or azathioprine. The immunosuppressive therapies are usually employed in patients with a high risk of progression, as characterized by proteinuria > 1.0 g/d and declining GFR (Cheng, Zhang et al. 2009, Boyd, Cheung et al. 2012, KDIGO 2012, Radhakrishnan and Cattran 2012, Barbour and Feehally 2017, Rodrigues, Haas et al. 2017). Recent trials have shown some benefit in proteinuria reduction with steroids in these patients, thought they are at high risk for developing significant complications like infections, metabolic derangements, osteoporosis, and diabetes mellitus with these immunosuppressive agents; thus, limiting the duration for which these drugs can be given to patients despite benefit from a renal perspective (Pozzi, Andrulli et al. 2004, Rauen, Eitner et al. 2015, Tesar, Troyanov et al. 2015, Lv, Zhang et al. 2017). Hence, there is a critical need for a safe and specific treatment for IgAN.

VIS649 has the potential to provide a significant advancement in the therapeutic approach to IgAN. It has a very specific mechanism of action in the form of APRIL inhibition, which plays a critical pathophysiological role in the production of a-g IgA<sub>1</sub> in patients with IgAN.

VIS649 has an attractive safety profile based on currently available data, including data from the first-in-human study, Study VIS649-101, in which no SAEs attributable to VIS649 were observed. It is anticipated that VIS649 will be used as a chronic therapy and will significantly improve the outcomes in patients with IgAN when compared to intermittent therapies like steroids that are currently being used to treat these patients.

#### 2.3.3 Overall Benefit: Risk Conclusion

Given the mechanism of action of VIS649 and data from a Phase 1 single-ascending dose study (Study VIS649-101) in healthy participants, it is expected that participants receiving VIS649 will

have a decline in the Immunoglobulin levels reduction, serum IgG thresholds for enrollment have been established so as to prevent the development of clinically significant hypogammaglobulinemia. In addition, studies in both healthy human participants and nonhuman primates have demonstrated that the ability to develop an IgG response to novel antigens and recall T-cell dependent antigen challenge is not significantly impaired. As mentioned earlier, there were no SAEs considered attributable to VIS649 in the Phase 1 single ascending dose study (VIS649-101), and in the nonhuman primate 6-month toxicology study, the no-adverse effect level for the antibody was the highest dose evaluated.

An independent data safety monitoring board (DSMB) for this study will be reviewing all available safety data, including unblinded Ig data and AEs on a periodic and ad-hoc basis as needed.

Given these encouraging preliminary data and the precautions built into the protocol, evaluation of the potential benefit of VIS649 in slowing or halting CKD progression in IgAN patients is warranted.

# 3. OBJECTIVES AND ENDPOINTS

Study objectives and endpoints are outlined in Table 3.

**Table 3:** Study Objectives and Endpoints

| Primary Safety Objective | Primary Safety Endpoint |
|---|---|
| To evaluate the safety and tolerability of multiple, monthly doses of VIS649 at each of 3 dosing levels, administered IV to IgAN participants over the course of 12 months as an add-on to SOC treatment with ACEI/ARB therapy, compared with saline placebo infusions as an add-on to SOC treatment with ACEI/ARB therapy | examinations |
| <b>Primary Efficacy Objective</b> | Primary Efficacy Endpoint |
| To evaluate the dose response of multiple, monthly doses of VIS649 on proteinuria at each of 3 dosing levels, administered IV to IgAN participants over the course of 12 months as an add-on to SOC treatment with ACEI/ARB therapy, compared with saline placebo infusions as an add-on to SOC treatment with ACEI/ARB therapy | Change from baseline in uPCR (measured on natural log scale from 24-hour urine collection or the intended 24-hour urine collection) at Month 12 (ie, approximately 30 days after the twelfth dose is administered) |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the effect of repeated doses of VIS649 at 3 dosing levels versus placebo on the following parameters: uPCR at Months 9 and 15 (ie, 4 months following the final [12th] monthly dose administration) 24-hour urine protein excretion at Month 9, 12, and 15 | <ul> <li>Change from baseline in uPCR (measured on natural log scale from 24-hour urine collection or the intended 24-hour urine collection) at Months 9 and 15</li> <li>Change from baseline in 24-hour urine protein excretion from baseline to</li> </ul> |
| <ul> <li>≥ 30% decline from baseline in uPCR at Months 9, 12, and 15.</li> </ul> | Months 9, 12, and 15 ○ Participants in each group achieving a ≥ 30% decline from baseline in uPCR at |
| <ul> <li>Clinical remission, defined as reduction in 24-hour urine protein excretion to &lt; 300 mg/day for at least 3 consecutive months.</li> </ul> | Months 9, 12, and 15 o Participants in each group achieving clinical remission |
| eGFR at Months 12 and 15 | • Change from baseline in eGFR at Months 12 and 15 |

- To evaluate the effect of repeated doses of VIS649 at each dosing level compared with placebo on the following PD parameters: IgA, IgG, and IgM concentrations
- To determine the PK profile of repeated dose of VIS649, at each dosing level
- To determine the PK/PD profile of VIS649, relating VIS649 PK parameters and biomarkers such as changes in IgA to changes in proteinuria and eGFR
- To screen for ADA responses

- Change from baseline in serum total IgA, IgG, and IgM concentrations at Months 9, 12, and 15
- Serum PK parameters
- Correlation of VIS649 PK parameters with changes in IgA, uPCR, and eGFR
- Serum ADA levels

# **Exploratory Objectives Exploratory Endpoints** • Explore the effect of VIS649 on urine albumin ı ı



Abbreviations: ACEI = angiotensin-converting enzyme inhibitor; ADA = anti-drug antibody; AE = adverse event; a-g IgA = aberrantly glycosylated immunoglobulin A; APRIL= A Proliferation Inducing Ligand; ARB = angiotensin receptor blocker; BAFF = B-cell activating factor; eGFR = estimated glomerular filtration rate; Ig = immunoglobulin; IgAN = immunoglobulin A nephropathy; IV = intravenous(ly); MEST = Mesangial cellularity, endocapillary proliferation, segmental sclerosis, tubular atrophy; PD = pharmacodynamic; PK = pharmacokinetic; SOC = standard of care; uACR = urinary albumin/creatinine ratio; uPCR = urinary protein/creatinine ratio.

#### 4. STUDY DESIGN

#### 4.1 Overall Design

This is a Phase 2 multicenter, randomized, double-blind, placebo-controlled, multiple-dose study to evaluate the safety and efficacy of IV administered VIS649 over a 12-month treatment course in participants with IgAN.

Participants will be enrolled from approximately 80 global sites in approximately 16 countries.

Screening evaluations (including physical examinations, vital signs, 12-lead electrocardiogram [ECG], safety laboratory testing [serum chemistry, hematology, urinalysis, serology, and pregnancy], and 24-hour urine collection) will take place during a 30-day time period prior to the first dose of study intervention.

To be eligible, participants should be on stable and maximally tolerated doses of either ACEI or ARB therapy, as per standard of care (SOC) and applicable guidelines, for at least 3 months. Participants must be on at least 50% of the recommended maximum dose of the ACEI or ARB to be considered as having adequate RAAS blockade.

Participants who are unable to tolerate ACEI/ARB therapy may be eligible for participation in the study if their overall management of IgAN, including BP control, is as per SOC and applicable guidelines.

Patient education regarding temporary cessation of ACEIs/ARBs during acute illness and resumption of these drugs after resolution of the acute illness will be as per local practice and SOC and this therapy will be resumed at the dose closest to the level at the time of randomization. During the course of the study, the doses of ACEIs or ARBs should not change; however, minor changes are allowed depending on the clinical situation. Control of BP should be as per SOC and applicable guidelines. Although additional anti-hypertensives can be used to control BP as per the Investigator's preference and local practice, combination of ACEIs and ARBs (or direct renin inhibitors) is prohibited and addition of mineral-corticoid receptor antagonists such as spironolactone or eplerenone should be avoided.

Enrolled participants must be adults, 18 years of age or older, with IgAN diagnosis confirmed by biopsy.

It is anticipated that most biopsies resulting in a diagnosis of IgAN will have been interpreted using the mesangial cellularity, endocapillary proliferation, segmental sclerosis, tubular atrophy (MEST) (Cattran et al, 2009) or MEST-C scoring system (Trimarchi, Barratt et al. 2017) from the Oxford classification of IgAN. Components of the MEST-C score include:

- M Mesangial hypercellularity, defined as more than 3 mesangial cells in any mesangial area of a glomerulus; a score of M0 indicates hypercellularity in < 50% of glomeruli and a score of M1 is for hypercellularity noted in ≥ 50% of glomeruli.
- E Endocapillary proliferation, defined as hypercellularity due to an increased number of cells within glomerular capillary lumina causing narrowing. E0 represents absence of hypercellularity; E1 is hypercellularity in any glomeruli.
- S Segmental glomerulosclerosis, defined as adhesion or sclerosis (obliteration of capillary lumina by matrix) in part of but not the whole glomerular tuft; S0 represents

absence of segmental glomerulosclerosis, S1 is presence of segmental glomerulosclerosis in any glomerulus.

- T Tubular atrophy/interstitial fibrosis, defined as the estimated percentage of cortical area showing tubular atrophy or interstitial fibrosis, whichever is greater; T0 is 0-25%; T1 is 25-50%; T2 is > 50% atrophy/interstitial fibrosis.
- C Crescents: C0 (no crescents), C1 (crescents in < 25% of glomeruli), and C2 (crescents in ≥ 25% of glomeruli).

A MEST-C score finding on kidney biopsy of T2 or C2 is exclusionary for this study. If the biopsy was not reported using the Oxford classification schema, the following findings are exclusionary: a) > 50% tubular atrophy, and/or b)  $\ge 25\%$  crescents.

Eligible participants must have sufficient proteinuria at Screening, defined as urine protein to creatinine ratio (uPCR)  $\geq 0.75$  g/g or 24-hour urine protein  $\geq 1.0$  g/d, as measured from a 24-hour urine collection (or an intended 24-hour urine collection). The proteinuria should be stable, as defined by a < 25% change when compared to values from  $\geq 3$  months ago (if available). If previous values are not available, or if the change from a prior value is  $\geq 25\%$ , a repeat measurement of proteinuria will be done after 15 days and the patient should fulfill the above proteinuria criteria to be eligible for randomization in the trial. Eligible participants must have an eGFR  $\geq 45$  mL/min/1.73 m², calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula (Levey, Stevens et al. 2009), before dosing on Day 1. The eGFR should be stable, as defined by a < 25% change when compared to values from  $\geq 3$  months ago (if available). If previous values are not available or if the change from a prior value is  $\geq 25\%$ , a repeat measurement of eGFR will be done after 15 days and the patient should fulfill the eGFR criteria to be eligible for randomization in the trial.

If the patient fulfills the proteinuria and eGFR criteria based on 2 measurements performed for each during the screening period, the second measurement (for each) will be considered as the baseline for analysis

Participants known to have chronic infectious diseases (eg, chronic sinusitis, chronic urinary tract infections, bronchiectasis) will be excluded. Participants in countries with high prevalence of tuberculosis may undergo appropriate investigations such as chest X-ray or interferon gamma-release assay, as deemed appropriate by the Investigator to rule out tuberculosis. Participants will be excluded from the study if they test positive for the screening serology markers listed in Table 7. Participants with a positive anti-hepatitis C virus (HCV) antibody test must undergo testing for HCV RNA; if HCV RNA is undetectable, the participant can be included in the study.

Participants must be vaccinated as per respective national guidelines and other relevant guidelines. Participants should continue to receive annual influenza vaccine and pneumococcal vaccine as per local guidelines.

The study will evaluate 3 dose levels of VIS649 (2, 4, and 8 mg/kg) versus placebo. A total of 144 participants will be randomized with equal allocation (1:1:1:1) across the 4 intervention groups (approximately 36 participants per group). Randomization will be stratified first by region (Japan vs rest-of-world). A target of twelve or more participants are planned to be randomized in Japan; these participants will be randomized with equal allocation and without

further stratification. The randomization for the rest-of-world will be stratified by screening uPCR ( $\leq 2.0 \text{ g/g vs} > 2.0 \text{ g/g}$ ).

VIS649 or placebo will be administered as twelve-monthly IV infusions starting on Day 1. Participants will return to the study center on Day 8 and then monthly through Month 12 for safety, PK and/or PD assessments. Participants will be encouraged to follow the schedule of visits for their monthly infusions as close to the prescribed interval as possible. If under special circumstances, a participant is unable to visit the study center within 7 days of the schedule infusion they may still be able to receive the infusion within the next 7 days, and this will be recorded as a protocol deviation. However, if there is any further delay, that dose should be skipped, and the participant should receive subsequent doses as per the schedule. The participant will not receive additional doses to make up for the missed dose.

Safety assessments will include review of AEs (including hypersensitivity reaction and anaphylactic reaction), physical examinations, injection site tolerability (including pain, irritation and tissue damage), clinical laboratory assessments (including biochemistry, hematology, and urinalysis), laboratory testing including serum Ig levels, vital sign measurements, and use of concomitant medications.

Participants will return to the study center on Month 15, approximately 120 days following the last dose of study intervention (Dose 12) for additional safety, PK, PD, and efficacy assessments. Participants discontinuing dosing prior to Dose 12 will attend an early termination visit at the time of dosing discontinuation and will be encouraged to attend the study visits as per schedule of assessments (Table 1).

An independent DSMB will review safety data at regular intervals (see Section 9.6).

It is anticipated that a roll-over extension study will be designed to enable longer term therapy for randomized participants. Further details will be provided in a separate protocol.

The total study duration for each participant (from screening to end-of-study [EOS]) will be up to 16 months (assuming 1 month for screening, 12 months for 12 monthly doses [through 30 days after the twelfth dose], and a 3-month safety follow-up).

# 4.2 Scientific Rationale for Study Design

This study is designed as a randomized, double-blind, placebo-controlled multiple-dose study to evaluate the safety and efficacy of intravenous (IV) administered VIS649 in IgAN participants over a 12-month intervention course.

Immunoglobulin A nephropathy is a chronic, slowly progressing disease. The underlying pathogenic factor in IgAN is the formation of a-g IgA<sub>1</sub>, which is attributed to a culmination of genetic and environmental factors in susceptible individuals. The hypoglycosylated hinge region of a-g IgA<sub>1</sub> presents as a novel antigen, against which IgG and IgA autoantibodies may be generated. This leads to formation of circulating IgG/a-g IgA<sub>1</sub> immune complexes, which are deposited (in part) in the mesangium of the glomerulus, inciting an inflammatory, nephritogenic response (Boyd, Cheung et al. 2012, Mestecky, Raska et al. 2013, Lv, Zhang et al. 2017). This manifests clinically as proteinuria, hematuria and decline in eGFR. High grade proteinuria (> 1.0 g/d) is a critical marker of progressive IgAN and remission of proteinuria is a crucial

therapeutic target in the management of IgAN (Donadio, Bergstralh et al. 2002, Reich, Troyanov et al. 2007, Nam, Kie et al. 2014, Inker, Mondal et al. 2016, Thompson, Carroll et al. 2019).

VIS649 inhibits the biological actions of APRIL and reduces the levels of IgA and other Ig. In patients with IgAN, it is hypothesized that this reduction in APRIL and a-g IgA<sub>1</sub> will reduce the deposition of circulating immunocomplexes in the glomerulus. This should lead to cessation of ongoing renal damage and lead to recovery of the damaged glomeruli, as reflected by a reduction in proteinuria.

Based on the PK/PD data from the Phase 1 single-ascending dose study (VIS649-101) and on simulation models, full therapeutic suppression of IgA through APRIL signaling inhibition will be achieved at 12 weeks, with the selected doses administered monthly. Considering the time-dependent and indirect effect of VIS649, a 12-month study intervention duration is deemed necessary to achieve therapeutic effect and assess for clinically relevant benefit of VIS649, as measured by reduction in proteinuria.

The primary efficacy endpoint will be the change from baseline in uPCR, at Month 12, 30 days after the twelfth dose of study intervention, as measured from a 24-hour urine collection. Studies have shown that in patients with IgAN, reduction of proteinuria leads to clinically relevant improvements like reduction in the rate of decline of eGFR and progression to ESRD.

In an analysis of data from the Toronto Glomerulonephritis Registry of 542 patients followed for a mean of 6.5 years (61% males, 50% whites, 23% Asians, with mean initial proteinuria 2.4 g/d, and creatinine clearance of 77 mL/min/1.73 m²), time-averaged proteinuria (defined as an average of the mean of the proteinuria measurements for every 6-month period) was the most important predictor of kidney function decline and risk of ESRD, independently of BP and use of renin-angiotensin blockers. If time-averaged proteinuria was maintained < 1 g/d, the 10-year risk of ESRD was 5%, versus 20% with a time-averaged proteinuria of 1–2 g/d, 40% with a time-averaged proteinuria of 2 to 3 g/d, and 60% with > 3 g/d (Reich, Troyanov et al. 2007).

This study highlights the primary importance of proteinuria reduction as a therapeutic target in the management of IgAN.

A comprehensive series of safety evaluations, including review of AEs (including hypersensitivity reaction and anaphylactic reaction), physical examinations, injection site tolerability (including pain, irritation and tissue damage), clinical laboratory assessments (including biochemistry, hematology, and urinalysis), laboratory testing including serum Ig levels, anti-drug antibody concentrations, vital sign measurements, and use of concomitant medications will be conducted to evaluate the safety profile of VIS649.

It is expected that VIS649 will result in obvious reductions in serum IgA, IgG, and IgM, which, if visible to the site or Sponsor, would effectively unblind treatment. Therefore, unblinded Ig data will only be available to designated unblinded personnel.

The DSMB will have access to the unblinded Ig data and will be responsible for monitoring Ig and AE data periodically (see Section 9.6).

#### 4.3 Justification for Dose

Three dose levels of monthly IV doses of VIS649 at 2, 4, and 8 mg/kg will be explored in this study.

Dose selection was informed by the totality of available nonclinical and clinical evidence, including safety margins from a 4-week and 6-month chronic toxicology study in cynomolgus monkeys and emerging data from the Phase 1 study using single doses from 0.5 to 12 mg/kg in healthy participants (Study VIS649-101).

Pharmacokinetic data from Study VIS649-101 demonstrate that there are no safety concerns when VIS649 levels are maintained above the effective concentration that inhibits APRIL and total serum IgA for  $\sim$ 2 and  $\sim$ 3 months, respectively, with single VIS649 doses of 6 and 12 mg/kg.

The anticipated pharmacologically active dose range in humans was evaluated using a PK/PD model based on data from Study VIS649-101. Simulation results predict that 2 mg/kg is the minimal dose that will achieve desired pharmacological activity with monthly dosing (Figure 2). Therefore, 2 mg/kg has been selected as the low dose for this study. It is possible, however, that higher APRIL levels and marked proteinuria in IgAN patients (versus healthy controls) could significantly accelerate VIS649 clearance. To mitigate this risk, 2 higher dose levels will be evaluated; 4 mg/kg and 8 mg/kg. Based on the PK/PD model simulations, VIS649 exposure after monthly 8 mg/kg doses is within the exposure range observed at 12 mg/kg in the Phase 1 single-dose study.



Figure 2: Simulated Percent Baseline Immunoglobulin A by Dose

Abbreviations: IgA = immunoglobulin A.

Note: Lines and shaded regions represent the median model prediction and model uncertainty (5<sup>th</sup> and 95<sup>th</sup> percentiles), respectively.

The results of Study VIS649-101 and of PK/PD model simulations and the safety coverage from the 6-month toxicology study all support the planned dosing strategy for the current study.

# **4.4** End of Study Definition

A participant is considered to have completed the study if he/she has completed all phases of the study including the EOS visit.

The end of the study is defined as the date of the last visit of the last participant in the study.
## 5. STUDY POPULATION

Prospective approval of protocol deviations to enrollment criteria, also known as protocol waivers or exemptions, is not permitted. Re-screening is typically not permitted, possible exceptions include re-testing of samples due to issues arising during shipping/storage/handling of samples. Re-screening of a participant may also be permitted if initial participation in the study was precluded due to an acute infection or an acute illness that subsequently resolved completely, and the participant is able to fulfill all study eligibility criteria.

#### 5.1 Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

- 1. Participant is a male or female ≥ 18 years of age at the time of signing the informed consent.
- 2. Participant must have biopsy-confirmed IgAN.
- 3. Participant medical records show they have been on stable and maximally tolerated doses of either ACEI or ARB, as per SOC and applicable guidelines, for at least 3 months preceding screening. Participants should be on at least 50% of the maximum recommended dose of these agents to be considered as having adequate RAAS blockade. Participants who are unable to tolerate ACEI/ARB therapy may be eligible for participation in the study if their overall management of IgAN, including BP control, is as per SOC and applicable guidelines.
- 4. Participants must have screening uPCR ≥ 0.75 g/g measured from a 24-hour urine (or an intended 24-hour urine sample) or 24-hour urine protein ≥ 1.0 g/d, as measured from 24-hour urine collection (or an intended 24-hour urine sample). The proteinuria should be stable, defined as < 25% change when compared to values from ≥ 3 months previously (if available).</p>
  - If previous values are not available or if the change from a prior value is > 25%, a repeat measurement of proteinuria will be done after 15 days and the participant should fulfill the above proteinuria criteria to be eligible for randomization in the study.
  - The proteinuria should be assessed when the participant is considered to be in a steady state with no recent heavy exercise, fever, or other potential issues that could impact the result.
- 5. Participants must have eGFR  $\geq$  45 mL/min/1.73 m<sup>2</sup>, calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula. The eGFR should be stable, as defined by a < 25% change when compared to values from  $\geq$  3 months previously (if available).
  - If previous values are not available or if the change from a prior value is > 25%, a repeat measurement of eGFR will be done after 15 days and the participant should fulfill the eGFR criteria to be eligible for randomization in the study.
  - The eGFR should be measured when the participant is considered to be in a steady state without recent changes in volume status, medications that could

impact the result (eg, nonsteroidal anti-inflammatory drugs [NSAIDs], aminoglycosides, co-trimoxazole) or changes in dietary protein intake.

- 6. Participant's serum Ig values must meet the criteria below:
  - $IgG: \ge 700 \text{ mg/dL}$
  - IgM:  $\geq 40 \text{ mg/dL}$
  - $IgA: \ge 70 \text{ mg/dL}$
- 7. Female participants of childbearing potential must have a negative serum pregnancy test prior to the first dose.
- 8. Participant is willing to adhere to contraceptive requirements outlined in Appendix 4.
- 9. Participant or a legally authorized representative is able to understand the purpose and risks of the study and is willing to give voluntary written informed consent as described in Appendix 1.

#### 5.2 Exclusion Criteria

Participants are excluded from the study if they meet any of the following criteria:

- 1. Participant has secondary forms of IgAN as defined by the treating physician (eg,, Henoch-Schönlein purpura, minimal change disease with IgA deposits, infection associated IgAN or IgAN associated with hepatic cirrhosis).
- 2. Participant has co-existing CKD, other than IgAN.
- 3. Participant has evidence of additional pathological findings in the kidney biopsy (eg, diabetic kidney disease, membranous nephropathy or lupus nephritis lupus). However, hypertensive vascular changes are acceptable.
- 4. Participant has kidney biopsy MEST or MEST-C score of T2 or C2 from the Oxford IgAN classification schema. If MEST-scoring was not performed, the presence of > 50% tubule-interstitial fibrosis or crescents in > 25% of glomeruli is exclusionary.
- 5. Participant has nephrotic syndrome, defined for this purpose as 24-hour urine protein > 3.5 g with concurrent hypoalbuminemia (serum albumin < 2.5 g/dL), hyperlipidemia (total cholesterol > 350 mg/dL) and edema.
- 6. Participant has received a solid organ transplant, including kidney.
- 7. Participant has received bone marrow or hematologic stem cell transplantation.
- 8. Participant is currently receiving systemic immunosuppression (excluding topical, ophthalmic, per rectum or inhaled corticosteroids).
- 9. Participant has received systemic steroids within the 12 weeks prior to initial screening.
- 10. Participant has received treatment with 2 or more systemic immunosuppressive agents within 2 years prior to initial screening.
- 11. Participant has chronic infectious diseases (eg, chronic urinary tract infection, chronic sinusitis, bronchiectasis, active pulmonary or systemic tuberculosis, chronic viral HCV or hepatitis B virus or HIV infection).

- 12. Participant has a known allergy or intolerance to any component of the study intervention.
- 13. Participant has acute infectious disease at the time of screening. Participants may be rescreened following resolution of acute infection (such as urinary tract infection or respiratory tract infection), provided there is no evidence of an immunosuppressive condition that predisposed the participant to this infection.
- 14. Participant has Type 1 diabetes.
- 15. Participant has uncontrolled Type 2 diabetes, as evidenced by a screening hemoglobin A1c value > 8%.
- 16. Participant has uncontrolled blood pressure (> 160 mm Hg systolic or > 110 mm Hg diastolic).
- 17. Participant has poorly compensated or controlled ischemic heart disease or cardiomyopathy, as judged by the Investigator.
- 18. Participant has chronic obstructive pulmonary disease (COPD) or asthma that has required systemic steroid therapy during the prior year. If COPD is present, severity must not exceed Global Initiative for Chronic Obstructive Lung Disease 1 (mild), defined as a forced 1-second expiratory volume (FEV<sub>1</sub>) > 80% of predicted.
- 19. Participant has known cirrhosis or liver dysfunction, defined as presence of coagulopathy, platelet count  $< 100,000/\mu L$  or alanine aminotransferase  $> 3 \times$  upper limit of normal (ULN).
- 20. Participant has history of chronic autoimmune neurodegenerative disorders (eg, multiple sclerosis).
- 21. Participant has active malignancy or is receiving chemotherapy for malignancy, except for nonmelanoma skin cancers and cervical carcinoma in situ. Participants with prior malignancy who have been documented to be cancer-free for ≥ 5 years may be enrolled.
- 22. Participant is planning or scheduled to undergo a tonsillectomy. Prior tonsillectomy is acceptable.
- 23. Participant enrolled in another investigational drug or device study within 3 months prior to initial screening.
- 24. Participant with a pre-existing illness other than those listed above that, in the opinion of the Investigator, would place the participant at increased risk through participation in this study.
- 25. Participant is unable to comply with study protocol procedures and/or study visit schedules.
- 26. Participant wit known or suspected alcohol or drug abuse that would compromise the safety or study participation and adherence of participant, in the opinion of the Investigator.

# 5.3 Lifestyle Considerations

Lifestyle recommendations applicable to IgAN patients such as, but not limited to, BP control, low-salt diet, low-protein diet, smoking cessation, weight reduction, and avoidance of nephrotoxic drugs such as NSAIDs will be followed as per local practice and guidelines.

## 5.4 Screen Failures

Screen failures are defined as participants who consent to participate in the clinical study but are not subsequently entered in the study. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants to meet the Consolidated Standards of Reporting Trials publishing requirements and to respond to queries from regulatory authorities. Minimal information includes demography, screen failure details, eligibility criteria, and any SAE.

#### 6. STUDY INTERVENTION

Study intervention is defined as any investigational intervention(s), marketed product(s), placebo, or medical device(s) intended to be administered to a study participant according to the study protocol.

# 6.1 Study Intervention(s) Administered

The study interventions to be administered under this protocol are detailed in Table 4.

VIS649 is for investigational use only and should only be used within the context of this study.

VIS649 will be administered as a mg/kg dosage determined by dose assigned at time of randomization. VIS649 will be administered IV over 1 hour, in a single, final volume 100 mL infusion in normal saline (0.9% NaCl), followed by a 25-mL saline flush. The dose of study intervention will be based on the Month 0 predose weight.

Placebo (0.9% NaCl) will be administered IV over 1 hour as a single 100 mL infusion, followed by a 25 mL saline flush.

Infusions should preferentially be administered to the participant's dominant arm.

**Table 4:** Study Interventions

| Study Arm | VIS649 | Placebo |
|---|---|---|
| Intervention Name | VIS649 | Placebo |
| Intervention Type | Drug (IMP) | Placebo (NIMP) |
| Dose Formulation | Solution | NaCl (normal saline solution) |
| Unit Dose Strength | VIS649 is formulated at a concentration of 25 mg/mL | 0.9% |
| Dosage Levels | 2.0, 4.0 and 8.0 mg/kg as a single, final volume of 100 mL | N/A |
| Dosing Frequency | Monthly for 12 months | Monthly for 12 months |
| Route of Administration | 1-hour IV infusion, followed by a 25-mL saline flush | 1-hour IV infusion, followed by a<br>25-mL saline flush |
| Use | Experimental | Placebo-comparator |
| Sourcing | Provided centrally by the Sponsor. | Supplies will be obtained locally |
| Packaging and Labeling | VIS649 will be supplied in vials containing a nominal volume of 10 mL and will be labeled according to local regulations | Per local supplies |
| Storage Conditions | VIS649 must be stored at a temperature between ≥ 2°C and ≤ 8°C and protected from light. Must be infused within 4 hours of reconstitution | Per package insert |

Abbreviations: ACEI = angiotensin-converting enzyme inhibitor; ARB = angiotensin receptor blocker; IMP = investigational medicinal product; IV = intravenous(ly); N/A = not applicable; NIMP = noninvestigational medicinal product; SOC = standard of care.

# 6.2 Preparation/Handling/Storage/Accountability

The required amount of VIS649 to be dosed will be diluted in normal saline up to a maximum total volume of 100 mL; for placebo participants, 100 mL of normal saline will be prepared. The length of the IV line will be set to a maximum volume of 25 mL, so that the 25-mL saline flush following administration will ensure all VIS649/placebo has been administered.

The VIS649/placebo infusion will be administered IV using a 0.20-µm in-line filter and will be controlled by a volumetric pump. Standard, uniform-length infusion lines will be used.

#### In addition:

- 1. The Investigator or designee must confirm appropriate temperature conditions have been maintained during transit for study intervention during transit to and storage in the investigational pharmacy, as well as post infusion solution preparations. Any deviations from Pharmacy Manual guidance are to be reported and resolved before use of the study intervention.
- 2. Only participants enrolled in the study may receive study intervention and only authorized site staff may supply or administer study intervention. All study intervention must be stored in a secure, environmentally controlled, and monitored (manual or automated) area in accordance with the labeled storage conditions with access limited to the Investigator and authorized site staff.
- 3. The Investigator, institution, or the head of the medical institution (where applicable) is responsible for study intervention accountability, reconciliation, and record maintenance (ie, receipt, reconciliation, and final disposition records).
- 4. Further guidance and information for the final disposition of unused study interventions are provided in the Study Reference Manual.

# 6.3 Measures to Minimize Bias: Randomization and Blinding

This study is double-blinded. An unblinded pharmacist will prepare study intervention doses for infusion. Participants, the Sponsor, the Investigator, and all other site study staff will be blinded to study intervention.

All eligible participants will be centrally assigned to randomized study intervention using an Interactive Voice/Web Response System (IVRS/IWRS). Before the study is initiated, the telephone number and call-in directions for the IVRS and/or the log in information and directions for the IWRS will be provided to each site.

Participants will be randomly assigned in a 1:1:1:1 allocation ratio to receive VIS649 at 2, 4, or 8 mg/kg, or placebo, with approximately 36 participants randomized to each intervention group. Randomization will be stratified first by region (Japan vs rest of world). A target of twelve or more participants are planned to be randomized at Japanese sites. Japanese participants will be randomized with equal allocation and without further stratification. Randomization for the rest of world will then be stratified by screening uPCR ( $\leq 2.0 \text{ g/g vs} > 2.0 \text{ g/g}$ ).

Each assignment will have a unique randomization number, assigned to eligible participants after the screening. Once a randomization number has been assigned via the IVRS/IWRS, it may not be reassigned.

In case of an emergency, the Investigator has the sole responsibility for determining if unblinding of a participants' intervention assignment is warranted. Participant safety must always be the first consideration in making such a determination. If the Investigator decides that unblinding is required for participant safety, the Investigator should make every effort to contact the Sponsor prior to unblinding a participant's intervention assignment unless this could delay emergency treatment of the participant. If a participant's intervention assignment is unblinded, the Sponsor must be notified within 24 hours after breaking the blind. The date and reason that the blind was broken must be recorded in the source documentation and electronic case report form (eCRF), as applicable.

Local laboratory testing such as Albumin:Globulin ratio (often tested as part of routine liver function panel) or serum protein electrophoresis, may reveal obvious reduction in the total globulin levels in participants receiving study intervention and will effectively unblind the participant, hence performing such investigations are prohibited, unless this has been discussed with the sponsors and if such investigations are deemed to be necessary for clinical management of the participant.

# **6.4** Study Intervention Compliance

Preparation of individual doses of study intervention will be confirmed by a second (unblinded) member of the study site pharmacy staff.

Participants will receive study intervention at the study center directly from the Investigator or designee, under medical supervision. The date and time of each dose administered in the clinic will be recorded in the source documents and recorded in the eCRF. The dose of study intervention and study participant identification will be confirmed at the time of dosing by a member of the study site staff other than the person administering the study intervention.

# 6.5 Concomitant Therapy

Any medication or vaccine (including over-the-counter and prescription medicines, vitamins, herbal supplements, fish oil, and NSAIDs) that the participant is receiving at the time of enrollment or receives during the study must be recorded along with:

- Reason for use
- Dates of administration including start and end dates
- Dosage information including dose and frequency

The Medical Monitor should be contacted if there are any questions regarding concomitant or prior therapy.

### 6.5.1 Concomitant Therapy to be Avoided

Participants should avoid using drugs that are relatively contraindicated in IgAN (eg, NSAIDs, aminoglycosides, co-trimoxazole) during the study, per local practice.

During conduct of the study, administration of systemic corticosteroids or other immunosuppressive therapy (for IgAN or other conditions) is prohibited due to the risk of over immune suppression due to overlapping actions of VIS649 and other immunosuppressive agents. If the Investigator believes that treatment with such therapy is required, and the potential benefits

outweigh the possible risks, the sponsor must be notified, as continued dosing with study intervention may, in this circumstance, be discontinued.

#### 6.6 Dose Modification

Participants will be encouraged to follow the schedule of visits for their monthly infusions as close to the prescribed interval as possible. If under special circumstances, a participant is unable to visit the study center within 7 days of the schedule infusion they may still be able to receive the infusion within the next 7 days, and this will be recorded as a protocol deviation. However, if there is any further delay, that dose should be skipped, and the participant should receive subsequent doses as per the schedule. The participant will not receive additional doses to make up for the missed dose.

There will be no other alterations from the dosing schedule outlined in Section 6.1.

# 6.7 Intervention after the End of the Study

It is anticipated that a rollover extension study will be designed to enable longer term therapy for randomized participants. Further details will be provided in a separate protocol.

# 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL

# 7.1 Discontinuation of Study Intervention Dosing

Participants have the right to discontinue study intervention or withdraw from the study at any time for any reason. Participants may withdraw or be withdrawn from study-related procedures and intervention for the following reasons:

- Withdrawal of consent
- Adverse event
- Protocol deviation
- Investigator decision
- Pregnancy (Appendix 4)
- Sponsor decision to terminate the study
- Loss to follow-up

In particular, study intervention should be discontinued if participants experience the following:

- Grade  $\geq 3$  infusion reaction such as severe anaphylaxis or cytokine release syndrome
- At the discretion of the Investigator, study intervention may be stopped if the participant has an unexplained decline of eGFR of > 30% sustained over 3 months that is not reversed after correction of all reversible factors such as volume depletion, NSAID, ACEI/ARB, other nephrotoxic drug use, or resolution of acute illness or infection.

All AEs should be followed until resolution or for a period of 30 days after the EOS, whichever is shorter (Section 8.3.1). If the participant withdrew because of an AE, every effort must be made to perform protocol-specified safety follow-up procedures.

If study intervention dosing is definitively discontinued, participants are encouraged to continue with assessments as per the schedule of assessments. At a minimum, if study participation is terminated by the participant or Investigator, the participant should complete all early termination assessments and will be encouraged to return for the EOS assessments outlined in Table 1. The primary reason for discontinuation should be recorded in the appropriate section of the eCRF.

#### 7.1.1 Temporary Discontinuation

Study intervention may be interrupted for up to 2 doses in participants who experience the following:

- Severe or intractable infection
- Acute severe illness or injury requiring hospitalization

#### 7.1.2 Rechallenge

VIS649 doses may be re-initiated (at the same dose) under the following conditions:

• If study intervention was interrupted due to acute illness or infection, study intervention can be re-initiated if the participant has recovered from the acute illness or infection, as determined by the Investigator.

# 7.2 Participant Discontinuation/Withdrawal from the Study

A participant may withdraw from the study at any time at his/her own request or may be withdrawn at any time at the discretion of the Investigator for safety, behavioral, compliance, or administrative reasons. This is expected to be uncommon.

At the time of discontinuing from the study, if possible, the participant should complete all ET assessments outlined in Table 1. The participant will be encouraged to attend an EOS visit approximately 120 days following the last dose of study intervention. The participant will be permanently discontinued both from the study intervention and from the study at that time.

If the participant withdraws consent for disclosure of future information, the Sponsor may retain and continue to use any data collected before such a withdrawal of consent.

If a participant withdraws from the study, he/she may request destruction of any samples taken and not tested, and the Investigator must document this in the site study records.

# 7.3 Lost to Follow-up

A participant will be considered lost to follow-up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site.

The following actions must be taken if a participant fails to return to the clinic for a required study visit:

- The site must attempt to contact the participant and reschedule the missed visit as soon as possible and counsel the participant on the importance of maintaining the assigned visit schedule and ascertain whether or not the participant wishes to and/or should continue in the study.
- Before a participant is deemed lost to follow up, the Investigator or designee must make every effort to regain contact with the participant (where possible, 3 telephone calls and, if necessary, a certified letter to the participant's last known mailing address or local equivalent methods). These contact attempts should be documented in the participant's medical record.
- Should the participant continue to be unreachable, he/she will be considered to have withdrawn from the study.

Discontinuation of specific sites or of the study as a whole are handled as part of Appendix 1.

# 8. STUDY ASSESSMENTS AND PROCEDURES

Study procedures and their timing are outlined in Table 1. Protocol waivers or exemptions are not allowed.

Immediate safety concerns should be discussed with the Sponsor immediately upon occurrence or awareness to determine if the participant should continue or discontinue study intervention.

Adherence to the study design requirements is essential and required for study conduct.

All screening evaluations must be completed and reviewed to confirm that potential participants meet all eligibility criteria. The Investigator will maintain a screening log to record details of all participants screened and to confirm eligibility or record reasons for screening failure, as applicable. A pathology report that confirms the IgAN diagnosis will be submitted with eCRFs.

Repeat or unscheduled samples may be taken for safety reasons or for technical issues with the samples.

# 8.1 Efficacy Assessments

# 8.1.1 Twenty-four-hour Urine Sample Collection

Twenty-four-hour urine collection for derivation of 24-hour urine volume, protein, albumin, and creatinine, uPCR, and uACR will be performed at the time points outlined in Table 1.

Participants will discard the first morning void and begin a 24-hour urine collection the day prior to the clinic visit. Care should be taken to avoid over-collection or under-collection of urine, however if this occurs, the sample may still be used to calculate the proteinuria and uPCR. On days of 24-hour urine collection (or the intended 24-hour urine collection), the uPCR sample will be collected from the 24-hour urine collection and routine urinalysis will be performed on a sample freshly voided during the clinic visit.

# 8.2 Safety Assessments

#### 8.2.1 Physical Examinations

A complete physical examination, to include assessments of the cardiovascular, respiratory, gastrointestinal and neurological systems will be completed at the screening and ET visit.

#### 8.2.2 Vital Signs

Vital sign measurements will be performed at the visits outlined in Table 1 and will include weight, temperature, pulse rate, respiratory rate, and systolic and diastolic BP. Height will be measured and recorded during Screening.

Vital signs measurements on dosing days will be recorded within 15 ( $\pm$ 5) minutes prior to the start of the infusion, every 15 minutes until the infusion is complete, and 60 minutes and 2 hours post infusion.

Systolic and diastolic BP and pulse measurements will be assessed while the participant is seated or supine with a completely automated device. Manual techniques will be used only if an automated device is not available. Blood pressure and pulse measurements should be preceded

by at least 5 minutes of rest for the participant in a quiet setting without distractions (eg, television, cell phones).

Vital signs should be to be collected before blood collection for laboratory tests, when possible, and before dosing with study intervention.

## 8.2.3 Electrocardiograms

A single 12-lead ECG, heart rate, and measures of PR, QRS, QT, and QTc intervals will be obtained at the screening visit. The 12-lead ECG should be conducted after 5 minutes in recumbence or semi-recumbency.

# 8.2.4 Clinical Safety Laboratory Assessments

Clinical laboratory evaluations for safety will be performed by a central laboratory whenever possible, however, local laboratory tests may be utilized for more urgent safety monitoring. Before starting the study, the Investigator will provide the Sponsor (or its designee) copies of all laboratory certifications and normal ranges for all laboratory assessments to be performed by that laboratory. Local laboratory assessments to make intervention-related decisions may be performed at all visits.

A list of clinical safety laboratory tests to be performed is provided in Appendix 2 and the timing for these assessments is provided in Table 1. All protocol-required laboratory assessments must be conducted in accordance with the laboratory manual. Details of laboratory tests to be conducted for assessment of VIS649 PK, PD, exploratory biomarkers, and immunogenicity are provided in Sections 8.5, 8.6, 8.8, and 8.9, respectively.

The Investigator must review the laboratory report, document this review, and record any clinically relevant changes occurring during the study in the AE section of the CRF. The laboratory reports must be filed with the source documents. Clinically significant abnormal laboratory findings are those which are not associated with the underlying disease, unless judged by the Investigator to be more severe than expected for the participant's condition.

All laboratory tests with values considered clinically significantly abnormal, with the exception of disease defining abnormalities such as eGFR and proteinuria considered to be a part of the natural history of IgAN, during participation in the study or within 30 days after the last dose of study intervention should be repeated until the values return to normal or baseline or are no longer considered clinically significant by the Investigator or medical monitor.

If such values do not return to normal/baseline within a period of time judged reasonable by the Investigator, the etiology should be identified, and the Sponsor notified.

# 8.3 Adverse Events and Serious Adverse Events

Adverse event and SAE definitions are provided in Appendix 3.

All AEs (serious and nonserious) reported by the participant must be recorded on the source documents and eCRF provided by the Sponsor. Medical terminology should be used for AE reporting. Adverse events should be reported as a single unifying diagnosis whenever possible or, in the absence of a unifying diagnosis, as individual signs or symptoms.

The Investigator and any qualified designees are responsible for detecting, documenting, and recording events that meet the definition of an AE or SAE and remain responsible for following up AEs that are serious, considered related to the study intervention or study procedures, or that caused the participant to discontinue the study intervention (see Section 7).

# 8.3.1 Time Period and Frequency for Collecting Adverse Event and Serious Adverse Event Information

All AEs and SAEs will be collected from the signing of the ICF until the EOS; AEs and SAEs that are ongoing at the EOS should be monitored until resolution or 30 days after EOS, whichever is shorter (see Section 1.3).

Medical occurrences that begin before the start of study intervention but after obtaining informed consent will be recorded on the Medical History/Current Medical Conditions section of the eCRF, not the AE section.

All SAEs will be recorded and reported to the Sponsor or designee immediately and under no circumstance should this exceed 24 hours, as indicated in Appendix 3. The Investigator will submit any updated SAE data to the Sponsor within 24 hours of it being available.

Investigators are not obligated to actively seek information about AEs or SAEs after conclusion of study participation. However, if the Investigator learns of any SAE, including a death, at any time after a participant has been discharged from the study, and he/she considers the event to be reasonably related to the study intervention or study participation, the Investigator must promptly notify the Sponsor.

## 8.3.2 Method of Detecting Adverse Events and Serious Adverse Events

The method of recording, evaluating, and assessing causality of AE and SAE and the procedures for completing and transmitting SAE reports are provided in Appendix 3.

Care will be taken not to introduce bias when detecting AEs and/or SAEs. Open-ended and nonleading verbal questioning of the participant is the preferred method to inquire about AE occurrences. For example, participants should be asked the nonleading question: "How have you felt since your last visit?"

**Exacerbation or disease progression** should be reported as an AE only if there are unusual or severe clinical features that were not present, or experienced earlier, or not expected based on the course of the condition.

In addition, the Sponsor must be notified immediately by telephone, fax, or e-mail of any immediately reportable events. Immediately reportable events (IRE) include the following:

- SAEs
- Pregnancies. Although normal pregnancy is not an AE, it will mandate study intervention
  discontinuation and must be reported on an IRE form and the Pregnancy Surveillance
  Form(s) to the Sponsor. Pregnancy will only be documented on the AE eCRF if there is
  an abnormality or complication. This includes pregnancy of the participant or the
  participant's partner

Adverse event, start date, end date, seriousness, severity, relationship to study intervention, action taken with study treatment and outcome will be recorded on the source documents and in

the eCRF. Special attention should be paid to recording hospitalization and concomitant medications.

#### 8.3.3 Follow-up of Adverse Events and Serious Adverse Events

Nonserious AEs that are identified at any time during the study must be recorded on the AE eCRF with the current status (ongoing or resolved/recovered) noted. All nonserious events (that are not IREs) that are ongoing at the last scheduled contact will be recorded as ongoing on the eCRF. For any AE having been identified throughout the study, additional relevant medical history information may be requested by the Sponsor during analysis to further ascertain causality (including, but not limited to, information such as risk-related behavior, family history and occupation).

After the initial AE/SAE report, the Investigator is required to proactively follow each participant at subsequent visits/contacts. All AEs and SAEs will be collected from the signing of the ICF until the EOS; AEs and SAEs that are ongoing at the EOS should be monitored until resolution, stabilization, until the event is otherwise explained, the participant is lost to follow-up or 30 days after EOS, whichever is shorter (Section 1.3).

Resolution means that the participant has returned to the baseline state of health and stabilized means that the Investigator does not expect any further improvement or worsening of the participant's condition. The Investigator will continue to report any significant follow-up information to the Sponsor up to the point the event has resolved or stabilized, or the participant is lost to follow-up, or has died.

Further information on follow-up procedures is provided in Appendix 3.

#### 8.3.4 Regulatory Reporting Requirements for Serious Adverse Events

Prompt notification by the Investigator to the Sponsor of a SAE is essential so that legal obligations and ethical responsibilities towards the safety of participants and the safety of a study intervention under clinical investigation are met.

The Sponsor has a legal responsibility to notify both the local regulatory authority and other regulatory agencies about the safety of a study intervention under clinical investigation. The Sponsor will comply with country-specific regulatory requirements relating to safety reporting to the regulatory authority, Institutional Review Boards (IRB)/Independent Ethics Committees (IEC), and Investigators.

Investigator safety reports must be prepared for suspected unexpected serious adverse reactions (SUSAR) according to local regulatory requirements and Sponsor policy and forwarded to Investigators as necessary.

An Investigator who receives an Investigator safety report describing a SAE or other specific safety information (eg, summary or listing of SAEs) from the Sponsor will review and then file it along with the Investigator's Brochure and will notify the IRB/IEC, if appropriate according to local requirements.

# 8.3.5 Pregnancy

Details of all pregnancies in female participants and female partners of male participants will be collected after the start of study intervention and until 90 days after the last dose of study intervention.

If a pregnancy is reported, the Investigator should inform the Sponsor within 24 hours of learning of the pregnancy and should follow the procedures outlined in Appendix 4.

Abnormal pregnancy outcomes (eg, spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) are considered SAEs.

## **8.4** Treatment of Overdose

Standard symptomatic support measures should be used in the case of excessive pharmacological effects or overdose. No antidotes are available.

#### 8.5 Pharmacokinetics

For all participants, serial blood samples will be drawn prior to each VIS649/placebo IV infusion and at the end of each infusion in order to determine circulating serum concentrations of VIS649, as specified in Table 1 and Table 5. Up to 60 participants (approximately 15 participants in each cohort) may have a more intensive PK and PD sampling schedule, as described in Table 5. Study participants who agree to participate in this more intensive PK and PD sample collection sub-study will sign an additional informed consent for this activity.

Instructions for the collection and handling of biological samples will be provided by the Sponsor in a separate laboratory manual. The actual date and time (24-hour clock time) of each sample will be recorded.

Samples collected for analyses of serum VIS649 concentration may also be used to evaluate safety or efficacy aspects related to concerns arising during or after the study.

Drug concentration information that may unblind the study will not be reported to investigative sites or blinded personnel until the study has been unblinded.

| | Day 1 | | Day 3 | Day 8 | Day 15 | |
|---|---|---|---|---|---|---|
| Time relative to infusion | Pre<br>infusion<br>(-30 min) | Post<br>infusion<br>(±15 min) | 2h<br>(±15 min) | 48h<br>(±1 day) | 168h<br>(±1 day) | 336h<br>(±3 days) |
| Month 0 | PK+Ig | PK only | PK only | PK only | PK+Ig | PK+Ig |
| Month 1 | PK+Ig | PK only | | | | PK+Ig |
| Month 2 | PK+Ig | PK only | | | | PK+Ig |
| Month 3 | PK+Ig | PK only | | | | PK+Ig |
| Months 4-10 | PK+Ig | PK only | | | | |
| Month 11 | PK+Ig | PK only | PK only | PK only | PK+Ig | PK+Ig |
| Month 12 | PK+Ig <sup>1</sup> | | | | | PK+Ig |
| Month 13 | PK+Ig <sup>1</sup> | | | | | PK+Ig |
| Month 14 | PK | +Ig <sup>1</sup> | | | | PK+Ig |
| Month 15 | PK | +Ig <sup>1</sup> | | | | |

Table 5: Pharmacokinetic and Serum Immunoglobulin Sampling Schedule

Abbreviations: IG = immunoglobulin; PK = pharmacokinetics.

# 8.6 Pharmacodynamics

Serial blood samples will be drawn in order to determine serum IgA, IgG, and IgM concentrations as well as the following analytes for exploratory PD endpoints

Up to 60 participants (approximately 15 participants in each cohort) will have a more intensive total serum IgA/IgM/IgG sampling schedule, as described in Table 5. Study participants who agree to participate in this more intensive sample collection sub-study will sign an additional informed consent for this activity.

It is expected that VIS649 will result in obvious reductions in serum IgA and IgM, which, if visible to site and Sponsor staff at the participant level, would effectively unblind treatment assignment. Participant level unblinded Ig data will not be available for review by the site or Sponsor staff. Unblinded Ig data will be routinely reviewed by the DSMB as part of the scheduled, if required, ad hoc safety reviews (see Section 9.6). Additional PK/PD summaries will be provided at an aggregate level in accordance with planned interim analyses (see Section 9.5).

#### 8.7 Genetics

A DNA sample will be collected to evaluate host DNA genetic markers related to IgAN susceptibility loci, the APRIL/B-cell activating factor pathway, and/or immunity in consenting subjects. Blood samples will be taken on Day 1 predose.

#### 8.8 Biomarkers

Collection of samples for other biomarker research is also part of this study. Participation is optional; a separate informed consent must be obtained. Participants who do not wish to

Note: postinfusion times are relative to the end of infusion.

No infusion on this date; therefore, only 1 sample to be obtained.



Samples may be stored in de-identified fashion for a maximum of 15 years (or according to local regulations) following the last participant's last visit for the study to enable further analysis of biomarker responses.

# 8.9 Immunogenicity Assessments

Antibodies to VIS649 will be evaluated in serum samples collected from all participants at the visits outlined in Table 1. Additionally, serum samples should also be collected at the final visit from participants who discontinued study intervention or were withdrawn from the study. These samples will be tested by the Sponsor or Sponsor's designee.

Serum samples will be screened for antibodies binding to VIS649 and the titer of confirmed positive samples will be reported. Other analyses may be performed to evaluate the stability of antibodies to VIS649 and/or further characterize the immunogenicity of VIS649.

The detection and characterization of antibodies to VIS649 will be performed using a validated assay method by or under the supervision of the Sponsor. All samples collected for detection of antibodies to VIS649 will also be evaluated for VIS649 serum concentration to enable interpretation of the antibody data. Antibodies may be further characterized and/or evaluated for their ability to neutralize VIS649 activity. Samples may be stored for a maximum of 15 years (or according to local regulations) following the last participant's last visit for the study at a facility selected by the Sponsor to enable further analysis of immune responses to VIS649. This analysis may be provided in a separate report.

# 8.10 Medical Resource Utilization and Health Economics

Not applicable

## 9. STATISTICAL CONSIDERATIONS

# 9.1 Statistical Hypothesis

The primary efficacy objective of this study is to evaluate the effect of VIS649 on proteinuria. The hypothesis that there is a VIS649-related dose response in the change from baseline in natural log uPCR at Month 12 versus placebo will be formally tested.

# 9.2 Sample Size Determination

A sample size of 144 participants, randomly assigned in a 1:1:1:1 schema to VIS649 2, 4, or 8 mg/kg, or placebo, would provide sufficient power at 80% to detect a significant linear dose response relationship given a standard deviation of 0.49, and an assumed difference in uPCR reduction, for instance 15%, 30%, and 45%, between VIS649 2, 4, or 8 mg/kg and placebo, respectively. The study-wide type I error rate is a 2-sided alpha of 0.05. This sample size would account for a dropout rate of ~20%.

# 9.3 Populations for Analyses

Populations for analysis in this study are defined in Table 6.

**Table 6:** Populations for Analysis

| Population | Description |
|---|---|
| ITT | All participants who are randomized; participants will be categorized by the intervention and dose they were randomized to receive. |
| mITT | All randomized participants who receive at least 1 dose of study intervention; participants will be categorized by the intervention and dose that they were randomized to receive. |
| Safety | All randomized participants who receive any amount of study intervention. Participants will be analyzed according to the intervention and dose they actually received. |
| PK/PD | All randomized participants who have at least 1 set of PK/PD measures taken. |
| Biomarker | All randomized participants who consented to participation in the biomarker sub-study. A separate consent process is required, as described in Section 8.8. |

Abbreviations: ITT = intent-to-treat; mITT = modified intent-to-treat; PD = pharmacodynamic(s); PK = pharmacokinetic(s).

Analysis of safety parameters will be performed on the Safety population. The Modified intent-to-treat (mITT) population will be the primary population for assessment of efficacy. The PK/PD population will be the primary population for PK/PD summaries. Analysis of biomarker data will be performed on the Biomarker population.

# 9.4 Statistical Analyses

The statistical analysis plan (SAP) will be finalized prior to database lock and it will include a more technical and detailed description of the statistical analyses described in this section. This section is a summary of the planned statistical analyses of the most important endpoints, including primary and key secondary endpoints.

#### 9.4.1 General considerations

All data collected will be documented using summary tables, figures, and/or participant data listings presented by intervention and dose group. For continuous variables, descriptive statistics (number [n], mean, geometric mean and coefficient of variation [%CV] as appropriate, median, standard deviation, minimum, and maximum) will be presented. For categorical variables, frequencies and percentages will be presented. As appropriate, a 95% CI will be presented. Graphical displays may be presented.

#### 9.4.2 Randomization and Stratification

Approximately 144 participants will be randomly assigned in a 1:1:1:1 ratio to study intervention or placebo, such that an estimated total of 36 participants are randomized per intervention group, with enrollment from approximately 80 global clinical sites in approximately 16 countries.

Randomization will be stratified first by region (Japan vs rest of world). A target of twelve or more participants are planned to be randomized at Japanese sites. Japanese participants will be randomized with equal allocation and without further stratification. Randomization for the rest of world will be stratified by screening uPCR ( $\leq 2.0 \text{ g/g}$  vs > 2.0 g/g).

#### 9.4.3 Participant Disposition

A tabulation of the disposition of participants will be presented by intervention group, including the number of participants randomized, number of participants mis-randomized, participant distribution for each stratification factor, number of participants treated, number of participants in each analysis population, reasons for study intervention discontinuation, and reasons for study discontinuation.

## 9.4.4 Participant Demographics

Demographic data based on the Safety population will be presented by intervention group and overall. Data to be tabulated will include sex, age, and race and ethnicity.

#### 9.4.5 Efficacy Analysis

Efficacy analyses will be performed on the mITT analysis population.

Additional detail for analysis methods will be described in the study SAP.

#### 9.4.5.1 Primary Endpoint

The primary efficacy outcome for this study is the change from baseline in uPCR on the natural log scale at Month 12. Dose response will be assessed using orthogonal contrasts. Sensitivity analysis will be performed using dose as a continuous covariate with associated linear, quadratic, and cubic terms.

In addition, to assess the dose response over time, a Mixed Model with Repeated Measurements (MMRM) including fixed class-effects of treatment, visit, strata factors, and treatment by visit interaction, and a fixed effect covariate of baseline uPCR on the natural log scale will be used.

An unstructured variance covariance matrix will be assumed, and liner, quadratic, and cubic dose responses will be assessed.

# 9.4.5.2 Secondary Endpoint(s)

Secondary efficacy endpoints will be summarized using descriptive statistics. In addition, comparisons between dose groups against placebo and between pooled dose groups against placebo will be performed using Analysis of Covariance or MMRM for continuous measures and logistic regression or generalized estimating equations for categorical variables.

Additional detail for analysis methods will be described in the SAP.

## 9.4.6 Safety Analyses

Safety will be assessed by evaluation of AEs (including hypersensitivity reaction and anaphylactic reaction), injection site tolerability (including irritation and tissue damage), clinical laboratory assessments (including biochemistry, hematology, and urinalysis), vital signs, and concomitant medications.

#### 9.4.7 Other Analyses

Analyses for PK, PK/PD, and antidrug antibodies (ADA) are described below. Additional detail on analysis of data, including analysis of other endpoints, will be described in the SAP.

## 9.4.7.1 Pharmacokinetic Analyses

VIS649 serum concentrations will be listed by participant and summary statistics, including arithmetic mean, geometric mean, standard deviation, %CV, median, and ranges, as appropriate, will be presented by intervention group. Summary graphs of mean concentration-time profiles by intervention group and ADA status will also be presented.

| For the subset of participants for whom intensive PK samples are collected, serum concentration |
|---|
| data will be analyzed . In addition, population PK methods |
| will be performed with NONMEM or equivalent |
| software. Additional analyses and summaries may be generated as appropriate. |
| Various techniques may be used to explore exposure-response |
| These techniques may include graphical and statistical methods, including the creation of |
| boxplots, spaghetti plots, histograms, and a variety of linear, nonlinear, or logistic regression |
| techniques and time-to-event methods. If appropriate, continuous independent variables will be |
| evaluated as such and as categorical variables, with participants grouped by exposure categories. |
| Additionally, population PK/PD modeling and simulation may be utilized to measure the |
| dynamic relationship between drug concentration, drug effect, and drug safety. |

#### 9.4.7.2 Anti-drug Antibodies

Presence vs absence of anti-VIS649 antibodies, anti-VIS649 antibody titers (including neutralizing antibody titers, if available), will be summarized by intervention group and time point using descriptive statistics.

# 9.5 Interim Analysis

In addition to five DSMB safety reviews (Section 9.6), three PK/Ig analyses and one interim efficacy analysis are planned:

- The first PK/Ig analysis will be performed when approximately 25% of participants have been randomized and have completed 3 months of study dosing. All the PK/Ig assessments will be performed by a separate, unblinded team. Summarized results will be made available to the study Sponsor for planning of future studies.
- The second PK/Ig analysis will be performed when approximately 20 participants have been randomized and have completed 9 months of study dosing. This analysis will be used to update previously developed population PK/PD models. Summarized results will be made available to the study Sponsor for planning of future studies.
- The third PK/Ig analysis will be performed when approximately 50% of the participants have been randomized and have completed 6 months of study dosing and approximately 20 participants have completed 12 months of study dosing. Summarized results will be made available to the study Sponsor for planning of future studies.
- An interim efficacy analysis will be performed at the time of the fourth scheduled DSMB meeting (when 50% of randomized participants have completed 6 months of study dosing and approximately 20 participants have completed 12 months of study dosing). Group-unblinded efficacy summaries (with individual participant treatment blinded) will be prepared for Sponsor review to inform future study design.
- The interim efficacy analysis will not include hypothesis testing and will be for the purpose of future study design and planning. The primary efficacy endpoint, change in proteinuria levels from baseline, will be analyzed. No modifications to this study protocol are planned based on results of the interim analyses.

# 9.6 Data Safety Monitoring Board

An independent DSMB will review unblinded safety data. The DSMB will meet at 5 scheduled data review meetings and on an ad hoc basis as needed. Details regarding the content and scope of safety assessments, as well as the governing of the DSMB, will be described in a separate DSMB charter. Data safety monitoring board meetings will be scheduled as the requirements in Table 7 are met.

| Table 7: | Scheduled Data | Safety Monitoring | <b>Board Reviews</b> |
|----------|----------------|-------------------|----------------------|
|----------|----------------|-------------------|----------------------|

| <b>Scheduled DSMB Review</b> | Number of Participants and Treatment Exposure |
|---|---|
| DSMB review #1 | The first scheduled meeting will occur after 12 participants have been randomized and have completed at least 3 months of dosing |
| DSMB review #2 | The second scheduled meeting will occur after 24 participants have been randomized and have completed at least 3 months of dosing |
| DSMB review #3 | The third scheduled meeting will occur after ~25% of participants have been randomized and have completed 3 months of dosing |


| DSMB review #4 | The fourth scheduled meeting will occur after ~50% of participants have been randomized and have completed 6 months of dosing and approximately 20 participants have completed 12 months of dosing |
|---|---|
| DSMB review #5 | The fifth scheduled meeting will occur after ~50% of participants have been randomized and have completed 12 months of dosing |

Abbreviations: DSMB = data safety monitoring board.

# 10. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

# 10.1 Appendix 1

# Regulatory, Ethical, and Study Oversight Considerations

## 10.1.1 Regulatory and Ethical Considerations

This study will be conducted in accordance with the protocol and with the following:

- Consensus ethical principles derived from international guidelines including the Declaration of Helsinki and Council for International Organizations of Medical Sciences (CIOMS) International Ethical Guidelines
- Applicable ICH Good Clinical Practice (GCP) Guidelines
- Applicable laws and regulations

The protocol, protocol amendments, ICF, Investigator Brochure, and other relevant documents (eg, advertisements) must be submitted to an IRB/IEC by the Investigator and reviewed and approved by the IRB/IEC before the study is initiated.

Any amendments to the protocol will require IRB/IEC approval before implementation of changes made to the study design, except for changes necessary to eliminate an immediate hazard to study participants.

The Investigator will be responsible for the following:

- Providing written summaries of the status of the study to the IRB/IEC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/IEC
- Notifying the IRB/IEC of SAEs or other significant safety findings as required by IRB/IEC procedures
- Providing oversight of the conduct of the study at the site and adherence to requirements of 21 CFR, ICH guidelines, the IRB/IEC, European regulation 536/2014 for clinical studies (if applicable), and all other applicable local regulations

#### **10.1.2** Financial Disclosure

All required information regarding financial certification or disclosure will be provided to the Sponsor for all investigators and sub investigators in accordance with the terms of the relevant regional regulation(s).

Informed consent will be freely obtained from all participants (or their guardian or legally acceptable representative, as applicable for local laws).

Each ICF will comply with the ICH (International Council for Harmonisation) Good Clinical Practice (GCP): Consolidated Guideline E6<sup>1</sup> and local regulatory requirements. The Investigator will ensure that the Sponsor reviews and authorizes any written site-specific ICF used in the study before submission to the IRB/IEC.

Investigators may discuss study availability and the possibility for entry with a potential participant without first obtaining consent. However, informed consent must be obtained and documented before initiation of any procedures that are performed solely for the purpose of determining eligibility for this study, including withdrawal from current medication(s).

Potential participants are free to refuse entry into the study, or withdraw from the study at any time, without justification, and there will be no consequences to their further care.

A separate and similar consent process will be followed for the optional blood samples for pharmacogenomic testing and future biospecimen research. Consent must be obtained before the blood sample is collected.

#### 10.1.3 Data Protection

All information generated in this study will be considered confidential and will not be disclosed to anyone not directly concerned with the study without the Sponsor's prior written permission. Participant confidentiality requirements of the region(s) where the study is conducted will be met. However, authorized regulatory officials and Sponsor personnel (or their representatives) may be allowed full access to inspect and copy the records, consistent with local requirements. All IMPs, participant bodily fluids, and/or other materials collected shall be used solely in accordance with this protocol, unless otherwise agreed to in writing by the Sponsor.

Participants will be identified only by unique participant ID in eCRF. If further participant identification is required, participants' full names may be made known to a regulatory agency or other authorized officials if necessary, subject to local regulations.

# 10.1.4 Dissemination of Clinical Study Data

This study will comply with the Clinical Trials Registration and Results Information Submission rule. As such, this study will be registered at ClinicalTrials.gov, and results information from this study will be submitted to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals. Data Quality Assurance

The accuracy and reliability of the study data will be assured by the selection of qualified Investigators and appropriate study centers, review of protocol procedures with the Investigator and associated personnel prior to the study, and by periodic monitoring visits by the Sponsor or designee.

Written instructions will be provided for the collection, preparation, and shipment of samples.

The Sponsor or its designee will review the EDC system for accuracy and completeness during (on-site) monitoring visits and after transmission to the Sponsor; any discrepancies will be resolved with the Investigator or designee, as appropriate. After upload of the data into the clinical study database, they will be verified for accuracy.

In accordance with Good Clinical Research Practice Guidelines and Recommendations, the Sponsor will be entitled to audit the facilities used in the clinical and laboratory parts of the study, as well as to access all the data files pertaining to the study. Similar procedures may also be conducted by agents of any regulatory body, either as part of a national GCP compliance program or to review the results of this study in support of a regulatory submission. The

Investigator should immediately notify the Sponsor if they have been contacted by a regulatory agency concerning an upcoming inspection.

#### **10.1.5** Source Documents

Source documents are defined as the results of original observations and activities of a clinical investigation. Source documents will include but are not limited to medical records, electronic data, screening logs, and recorded data from automated instruments. All source documents pertaining to this study will be maintained by the Investigators and made available for direct inspection by authorized persons.

Investigator(s)/institution(s) will permit study -related monitoring, audits, [IRB/IEC/EC] review, and regulatory inspection(s) by providing direct access to source data/documents by authorized persons as defined in the ICF. In all cases, participant confidentiality must be maintained in accordance with local regulatory requirements.

## 10.1.6 Study and Site Start and Closure

Study site participation may be discontinued if the Sponsor or its designee, the Investigator, or the ethical review board (ERB) of the study site judges it necessary for medical, safety, regulatory, or other reasons consistent with applicable laws, regulations, and GCP. 10.3.2.

The study will be discontinued if the Sponsor or its designee judges it necessary for medical, safety, regulatory, or other reasons consistent with applicable laws, regulations, and GCP.

## **10.1.7** Publication Policy

The publication policy for the study will be documented in the agreement between the Sponsor and the Investigator. Authorship for any Visterra-Sponsored publications resulting from the conduct of this study will be based on International Committee of Medical Journal Editors (ICMJE) authorship criteria (http://www.icmje.org/recommendations). According to ICMJE guidelines, one may be considered an author only if the following criteria are met:

- 1. Substantial contributions to the conception or design of the work; or the acquisition, analysis, or interpretation of data for the work; AND
- 2. Drafting the work or revising it critically for important intellectual content; AND
- 3. Final approval of the version to be published; AND
- 4. Agreement to be accountable for all aspects of the work in ensuring that questions related to the accuracy or integrity of any part of the work are appropriately investigated and resolved.

All authors must meet the above criteria, and all who qualify for authorship based on the above criteria should be listed as authors.

# 10.2 Appendix 2

# **Clinical Laboratory Tests**

Table 7 provides a list of laboratory tests to be evaluated by the Investigator.

The tests detailed in Table 7 will be performed by the central laboratory.

Local laboratory results are only required in the event that the central laboratory results are not available in time for either study intervention administration and/or response evaluation. If a local sample is required, it is important that the sample for central analysis is obtained at the same time. Additionally, if the local laboratory results are used to make either a study intervention decision or response evaluation, the results must be entered into the eCRF. Local lab results will not be acceptable for qualifying a participant for the study.

Additional tests may be performed at any time during the study as determined necessary by the Investigator or required by local regulations.

**Table 8: Protocol-Required Safety Laboratory Assessments** 

| Serology (screening only) | HBsAg, anti-HBc (IgG and IgM) antibody, anti-HCV antibody, HIV |
|---|---|
| Hematology | Hemoglobin, RBC, WBC with differential (including absolute neutrophil count), and platelet count |
| Serum chemistry | Sodium, potassium, BUN, bicarbonate (venous), creatinine, calcium, chloride, magnesium, phosphorus, albumin, AST, ALT, ALP, total bilirubin (direct bilirubin if total > ULN), total cholesterol and triglycerides. |
| Urinalysis | Color and appearance; pH, specific gravity, ketones, protein, glucose, bilirubin, nitrite, urobilinogen, and occult blood by dipstick |
| Pregnancy (females only) | Serum β-hCG (screening only) Urine β-hCG (all other visits) |

Abbreviations: ALP = alkaline phosphatase; ALT = alanine aminotransferase; AST = aspartate aminotransferase;  $\beta$ -hCG =  $\beta$ -human chorionic gonadotropin; BUN = blood urea nitrogen; HBc = hepatitis B core; HBsAg = hepatitis B surface antigen; HCV = hepatitis C virus; HIV = human immunodeficiency virus; RBC = red blood cell; ULN = upper limit of normal; WBC = white blood cell.

Note: eGFR will be calculated from Serum creatinine by the CKD-EPI formula, which is as follows: eGFR =141 x min  $(S_{Cr}/\kappa, 1)^{\alpha}$  x max $(S_{Cr}/\kappa, 1)^{-1.209}$  x 0.993 Age x 1.018 [if female] x 1.159 [if Black]  $\kappa$  = 0.7 (females) or 0.9 (males),  $\alpha$  = -0.329 (females) or -0.411 (males), min = indicates the minimum of  $S_{Cr}/\kappa$  or 1, max = indicates the maximum of  $S_{Cr}/\kappa$  or 1. Investigators must document their review of each laboratory safety report.

Laboratory results that could unblind the study (eg, Ig) will not be reported to investigative sites or other blinded personnel until the study has been unblinded.

# 10.3 Appendix 3

# Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting

## 10.3.1 Definition of Adverse Event and Adverse Reaction

#### Adverse Event Definition

- An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
- An AE would not include information recorded as medical history at screening for preplanned procedures for which the underlying condition was known and no worsening occurred.
- NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention.
- Treatment-emergent AEs (TEAEs) are defined as AEs with an onset date on or after the start of
  study intervention. In more detail, TEAEs are all adverse events which started after start of
  study intervention; or if the event was continuous from baseline and was worsening, serious,
  study intervention-related, or resulted in death, discontinuation, interruption or reduction of
  study intervention dose.
- A suspected adverse reaction is any AE for which there is a reasonable possibility that the
  study intervention caused the AE. For the purpose of Investigational New Drug safety
  reporting, "reasonable possibility" means there is evidence to suggest a causal relationship
  between the study intervention and the AE. Suspected adverse reaction implies a lesser degree
  of certainty about causality.

#### **Events Meeting the Adverse Event Definition**

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or other safety assessments (eg, ECG, radiological scans, vital signs measurements), including those that worsen from baseline, considered clinically significant in the medical and scientific judgment of the Investigator (ie, not related to progression of underlying disease). It is the Investigator's responsibility to review the results of laboratory tests for each individual participant as they become available. This review will be documented by the Investigator's dated signature on the laboratory report. The Investigator may repeat the laboratory test or request additional tests to verify the results of the original laboratory tests.
- Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition.
- New conditions detected or diagnosed after study intervention administration even though it
  may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study intervention
  or a concomitant medication. Overdose per se will not be reported as an AE/SAE unless it is an
  intentional overdose taken with possible suicidal/self-harming intent. Such overdoses should be
  reported regardless of sequelae.

## Events NOT Meeting the Adverse Event Definition

- Any clinically significant abnormal laboratory findings or other abnormal safety assessments
  which are associated with the underlying disease, unless judged by the Investigator to be more
  severe than expected for the participant's condition.
- The disease/disorder being studied or expected progression, signs, or symptoms of the disease/disorder being studied, unless more severe than expected for the participant's condition.
- Medical or surgical procedure (eg, endoscopy, appendectomy): the condition that leads to the procedure is the AE.
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).
- Anticipated day-to-day fluctuations of pre-existing disease(s) or condition(s) present or detected at the start of the study that do not worsen.

#### 10.3.2 Definition of Serious Adverse Event

If an event is not an AE per the definition above, then it cannot be an SAE even if serious conditions are met (eg, hospitalization for signs/symptoms of the disease under study, death due to progression of disease).

#### A Serious Adverse Event Is Defined as Any Untoward Medical Occurrence That, at Any Dose:

#### Results in death

#### • Is life-threatening

The term 'life-threatening' in the definition of 'serious' refers to an event in which the participant was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, if it were more severe.

#### • Requires inpatient hospitalization or prolongation of existing hospitalization

In general, hospitalization signifies that the participant has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred or was necessary, the AE should be considered serious.

Hospitalization itself should not be reported as an SAE; whenever possible the reason for the hospitalization should be reported.

Hospitalizations or prolonged hospitalizations for social admissions (ie, those required for reasons of convenience or other nonmedical need) are not considered SAEs.

Hospitalization for elective treatment of a pre-existing condition that did not worsen from baseline is not considered an AE.

#### Results in persistent disability/incapacity

The term disability means a substantial disruption of a person's ability to conduct normal life functions.

This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (eg, sprained ankle) which may interfere with or prevent everyday life functions but do not constitute a substantial disruption.

#### • Is a congenital anomaly/birth defect

#### Other situations:

Medical or scientific judgment should be exercised in deciding whether SAE reporting is appropriate in other situations such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition. These events should usually be considered serious.

Examples of such events include invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

#### 10.3.3 Recording and Follow-Up of Adverse Event and/or Serious Adverse Event

#### Adverse Event and Serious Adverse Event Recording

- When an AE/SAE occurs, it is the responsibility of the Investigator to review all
  documentation (eg, hospital progress notes, laboratory reports, diagnostics reports) related to
  the event.
- The Investigator will then record all relevant AE/SAE information in the eCRF.
- It is not acceptable for the Investigator to send photocopies of the participant's medical records in lieu of completion of the AE/SAE CRF page.
- There may be instances when copies of medical records for certain cases are requested. In this
  case, all participant identifiers, with the exception of the participant number, will be redacted
  on the copies of the medical records before submission.
- The Investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. Whenever possible, the diagnosis (not the individual signs/symptoms) will be documented as the AE/SAE.

#### Assessment of Intensity

The Investigator will make an assessment of intensity for each AE and SAE reported during the study and assign it to one of the following categories:

- Mild: An event that is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities.
- Moderate: An event that causes sufficient discomfort and interferes with normal everyday activities.
- Severe: An event that prevents normal everyday activities. An AE that is assessed as severe should not be confused with a SAE. Severe is a category utilized for rating the intensity of an event; and both AEs and SAEs can be assessed as severe.

An event is defined as 'serious' when it meets at least one of the predefined outcomes as described in the definition of an SAE, NOT when it is rated as severe.

#### **Assessment of Causality**

The Investigator is obligated to assess the relationship between study intervention and each occurrence of each AE/SAE. Assessment of causal relationship of an AE to the study intervention is defined as follows:

 Related: There is a reasonable possibility of a temporal and causal relationship between study intervention and the AE.  Not Related: There is no temporal or causal relationship between study intervention and the AE.

The Investigator will use clinical judgment to determine the relationship. Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study intervention administration will be considered and investigated. The Investigator will also consult the Investigator's Brochure (IB) and/or Product Information, for marketed products, in his/her assessment.

For each AE/SAE, the Investigator **must** document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of causality. There may be situations in which an SAE has occurred and the Investigator has minimal information to include in the initial report. However, it is very important that the Investigator always make an assessment of causality for every event before the initial transmission of the SAE data.

The Investigator may change his/her opinion of causality in light of follow-up information and send a SAE follow-up report with the updated causality assessment.

The causality assessment is one of the criteria used when determining regulatory reporting requirements.

#### Follow-up of Adverse Events and Serious Adverse Events

The Investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as medically indicated to elucidate the nature and/or causality of the AE or SAE as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other health care professionals.

New or updated information will be recorded in the originally completed eCRF.

The Investigator will submit any updated SAE data to the Sponsor within 24 hours of receipt of the information

#### 10.3.4 Reporting of Serious Adverse Events

#### SAE Reporting via an Electronic Data Collection Tool

- The primary mechanism for reporting an SAE will be the electronic data collection tool.
- If the electronic system is unavailable, then the site will use the paper SAE data collection tool (see next section) in order to report the event within 24 hours.
- The site will enter the SAE data into the electronic system as soon as it becomes available.
- After the study is completed at a given site, the electronic data collection tool will be taken offline to prevent the entry of new data or changes to existing data.
- If a site receives a report of a new SAE from a study participant or receives updated data on a
  previously reported SAE after the electronic data collection tool has been taken offline, then
  the site can report this information on a paper SAE form or to the Medical Monitor by
  telephone.



# 10.4 Appendix 4

# Contraceptive Guidance and Collection of Pregnancy Information

#### 10.4.1 Definitions

## Woman of Childbearing Potential (WOCBP)

A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile (see below).

If fertility is unclear (eg, amenorrhea in adolescents or athletes) and a menstrual cycle cannot be confirmed before first dose of study intervention, additional evaluation should be considered.

Women in the following categories are not considered WOCBP:

- 1. Premenarchal
- 2. Premenopausal female with 1 of the following:
  - Documented hysterectomy
  - Documented bilateral salpingectomy
  - Documented bilateral oophorectomy

For individuals with permanent infertility due to an alternate medical cause other than the above (eg, mullerian agenesis, androgen insensitivity), Investigator discretion should be applied to determining study entry.

Note: Documentation can come from site personnel review of the participant's medical records, medical examination, or medical history interview.

- 3. Postmenopausal female
  - A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
    - A high follicle-stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy (HRT). However, in the absence of 12 months of amenorrhea, confirmation with more than one FSH measurement is required.
    - Females on HRT and whose menopausal status is in doubt will be required to use one of the nonestrogen hormonal highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrollment.

# 10.4.2 Contraception Guidance

Women of childbearing potential must use a medically acceptable form of birth control (hormonal contraception, diaphragm with spermicide, condom with spermicide, intrauterine device, or partner with vasectomy) for at least 28 days prior to first study intervention and agree to continue to use a medically acceptable form of birth control (as described) through 90 days

after the last dose of study intervention. Alternatively, a reported history of abstinence beginning at least 28 days prior to study intervention dosing, with agreement to continue abstinence through 90 days after the last dose of study intervention are required. Women of childbearing potential must also have a negative serum beta human chorionic gonadotropin ( $\beta$ -hCG) pregnancy test at screening and a negative urine  $\beta$ -hCG pregnancy test prior to the first study intervention on Day 0. Female participants must also agree not to donate eggs/bank eggs for the duration of their participation in the study.

Male participants and/or his partner must use a highly effective form of contraception (ie, double-barrier as described above, have had a vasectomy, or have a female partner of nonchildbearing potential) from date of first study dose through 90 days after the last dose of study intervention. Following the first dose of study intervention, male participants must also agree to not donate sperm through 90 days after the last dose of study intervention.

## 10.4.3 Collection of Pregnancy Information

## Male participants with partners who become pregnant

- The Investigator will attempt to collect pregnancy information on any male participant's female partner who becomes pregnant while the male participant is in this study. This applies only to male participants who receive study intervention.
- After obtaining the necessary signed informed consent from the pregnant female partner directly, the Investigator will record pregnancy information on the appropriate form and submit it to the Sponsor within 24 hours of learning of the partner's pregnancy. The female partner will also be followed to determine the outcome of the pregnancy. Information on the status of the mother and child will be forwarded to the Sponsor. Generally, the follow-up will be no longer than 6 to 8 weeks following the estimated delivery date. Any termination of the pregnancy will be reported regardless of fetal status (presence or absence of anomalies) or indication for the procedure.

#### Female participants who become pregnant

- The Investigator will collect pregnancy information on any female participant who becomes pregnant while participating in this study. The initial information will be recorded on the appropriate form and submitted to the Sponsor within 24 hours of learning of a participant's pregnancy.
- The participant will be followed to determine the outcome of the pregnancy. The Investigator will collect follow-up information on the participant and the neonate and the information will be forwarded to the Sponsor. Generally, follow-up will not be required for longer than 6 to 8 weeks beyond the estimated delivery date. Any termination of the pregnancy will be reported regardless of fetal status (presence or absence of anomalies) or indication for the procedure.
- While pregnancy itself is not considered to be an AE or SAE, any pregnancy complication or elective termination of a pregnancy for medical reasons will be reported as an AE or SAE.

- A spontaneous abortion (occurring at < 22 weeks gestational age) or still birth (occurring at > 22 weeks gestational age) is always considered to be an SAE and will be reported as such.
- Any poststudy pregnancy related SAE considered reasonably related to the study intervention by the Investigator will be reported to the Sponsor as described in Section 8.3.4. While the Investigator is not obligated to actively seek this information in former study participants, he or she may learn of an SAE through spontaneous reporting.
- Any female participant who becomes pregnant while participating in the study will discontinue study intervention.

# 10.5 Appendix 5

# **Abbreviations**

| Abbreviation | Definition |
|------------------|-------------------------------------------------------|
| ACEI | Angiotensin-converting enzyme inhibitor |
| ADA | Antidrug antibody |
| AE | Adverse event |
| a-g | Aberrantly glycosylated |
| AKI | Acute kidney injury |
| ALT | Alanine aminotransferase |
| APRIL | Cytokine A proliferation inducing ligand |
| ARB | Angiotensin receptor blocker |
| AST | Aspartate aminotransferase |
| AUC | Area under the serum concentration versus -time curve |
| β-hCG | Beta human chorionic gonadotropin |
| BCMA | B-cell maturation antigen |
| BP | Blood pressure |
| CKD | Chronic kidney disease |
| CKD-EPI | Chronic Kidney Disease Epidemiology Collaboration |
| $C_{\text{max}}$ | Maximum serum concentration |
| COPD | Chronic obstructive pulmonary disease |
| %CV | Coefficient of variation |
| DSMB | Data safety monitoring board |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| eGFR | Estimated glomerular filtration rate |
| EOS | End-of-study |
| ESRD | End-stage renal disease |
| FSH | Follicle-stimulating hormone |
| GCP | Good Clinical Practice |
| GFR | Glomerular filtration rate |
| HCV | Hepatitis C virus |
| HRT | Hormone-replacement therapy |
| IEC | Independent Ethics Committee |
| Ig | Immunoglobulin |

**Abbreviation Definition** 

IgA/G/M Immunoglobulin A/G/M

IgAN Immunoglobulin A nephropathy

IRB Institutional Review Board

IRE Immediately reportable event

IV Intravenous

IVRS/IWRS Interactive voice/web response system

LS Least-squares

mAb Monoclonal antibody

MEST-C Mesangial cellularity, Endocapillary proliferation, Segmental sclerosis,

Tubular atrophy, Crescents

mITT Modified intent-to-treat

MMRM Mixed Model Repeated Measurement
NSAID Nonsteroidal anti-inflammatory drug

PD Pharmacodynamic(s)
PK Pharmacokinetic(s)

RAAS Renin-angiotensin-aldosterone system

SAE Serious Adverse Event
SAP Statistical Analysis Plan

SOC Standard of care

SUSAR Suspected unexpected serious adverse reaction

TACI Transmembrane activator and CAML interactor

Td Tetanus and diphtheria
ULN Upper limit of normal

uPCR Urine protein to creatinine ratio
WOCBP Woman of childbearing potential

## 11. REFERENCES

Ballow, M. (2002). "Primary immunodeficiency disorders: antibody deficiency." <u>J Allergy Clin Immunol</u> **109**(4): 581-591.

Barbour, S. and J. Feehally (2017). "An update on the treatment of IgA nephropathy." <u>Curr Opin Nephrol Hypertens</u> **26**(4): 319-326.

Berthoux, F., H. Suzuki, L. Thibaudin, H. Yanagawa, N. Maillard, C. Mariat, Y. Tomino, B. A. Julian and J. Novak (2012). "Autoantibodies targeting galactose-deficient IgA1 associate with progression of IgA nephropathy." <u>J Am Soc Nephrol</u> **23**(9): 1579-1587.

Bossen, C., T. G. Cachero, A. Tardivel, K. Ingold, L. Willen, M. Dobles, M. L. Scott, A. Maquelin, E. Belnoue, C. A. Siegrist, S. Chevrier, H. Acha-Orbea, H. Leung, F. Mackay, J. Tschopp and P. Schneider (2008). "TACI, unlike BAFF-R, is solely activated by oligomeric BAFF and APRIL to support survival of activated B cells and plasmablasts." <u>Blood</u> **111**(3): 1004-1012.

Boyd, J. K., C. K. Cheung, K. Molyneux, J. Feehally and J. Barratt (2012). "An update on the pathogenesis and treatment of IgA nephropathy." <u>Kidney Int</u> **81**(9): 833-843.

Castigli, E., S. Scott, F. Dedeoglu, P. Bryce, H. Jabara, A. K. Bhan, E. Mizoguchi and R. S. Geha (2004). "Impaired IgA class switching in APRIL-deficient mice." <u>Proc Natl Acad Sci U S</u> A **101**(11): 3903-3908.

Cheng, J., W. Zhang, X. H. Zhang, Q. He, X. J. Tao and J. H. Chen (2009). "ACEI/ARB therapy for IgA nephropathy: a meta analysis of randomised controlled trials." <u>Int J Clin Pract</u> **63**(6): 880-888.

Donadio, J. V., E. J. Bergstralh, J. P. Grande and D. M. Rademcher (2002). "Proteinuria patterns and their association with subsequent end-stage renal disease in IgA nephropathy." <u>Nephrology</u> Dialysis Transplantation 17(7): 1197-1203.

Endo, T., M. Nishio, T. Enzler, H. B. Cottam, T. Fukuda, D. F. James, M. Karin and T. J. Kipps (2007). "BAFF and APRIL support chronic lymphocytic leukemia B-cell survival through activation of the canonical NF-kappaB pathway." <u>Blood</u> **109**(2): 703-710.

Fadlallah, J., H. El Kafsi, D. Sterlin, C. Juste, C. Parizot, K. Dorgham, G. Autaa, D. Gouas, M. Almeida, P. Lepage, N. Pons, E. Le Chatelier, F. Levenez, S. Kennedy, N. Galleron, J. P. de Barros, M. Malphettes, L. Galicier, D. Boutboul, A. Mathian, M. Miyara, E. Oksenhendler, Z. Amoura, J. Dore, C. Fieschi, S. D. Ehrlich, M. Larsen and G. Gorochov (2018). "Microbial ecology perturbation in human IgA deficiency." Sci Transl Med 10(439).

Floege, J., I. C. Moura and M. R. Daha (2014). "New insights into the pathogenesis of IgA nephropathy." <u>Semin Immunopathol</u> **36**(4): 431-442.

Furst, D. E. (2009). "Serum immunoglobulins and risk of infection: how low can you go?" Semin Arthritis Rheum **39**(1): 18-29.

- Han, S. S., S. H. Yang, M. Choi, H. R. Kim, K. Kim, S. Lee, K. C. Moon, J. Y. Kim, H. Lee, J. P. Lee, J. Y. Jung, S. Kim, K. W. Joo, C. S. Lim, S. W. Kang, Y. S. Kim and D. K. Kim (2016). "The Role of TNF Superfamily Member 13 in the Progression of IgA Nephropathy." <u>J Am Soc Nephrol</u> **27**(11): 3430-3439.
- Hastings, M. C., Z. Bursac, B. A. Julian, E. Villa Baca, J. Featherston, S. Y. Woodford, L. Bailey and R. J. Wyatt (2017). "Life Expectancy for Patients From the Southeastern United States With IgA Nephropathy." <u>Kidney international reports</u> **3**(1): 99-104.
- Inker, L. A., H. Mondal, T. Greene, T. Masaschi, F. Locatelli, F. P. Schena, R. Katafuchi, G. B. Appel, B. D. Maes, P. K. Li, M. Praga, L. Del Vecchio, S. Andrulli, C. Manno, E. Gutierrez, A. Mercer, K. J. Carroll, C. H. Schmid and A. S. Levey (2016). "Early Change in Urine Protein as a Surrogate End Point in Studies of IgA Nephropathy: An Individual-Patient Meta-analysis." <u>Am J Kidney Dis</u> **68**(3): 392-401.
- Janssen, L. M. A., T. Macken, M. C. W. Creemers, J. F. M. Pruijt, J. J. J. Eijk and E. de Vries (2018). "Truly selective primary IgM deficiency is probably very rare." <u>Clin Exp Immunol</u> **191**(2): 203-211.
- Jarrick, S., S. Lundberg, A. Welander, J. J. Carrero, J. Hoijer, M. Bottai and J. F. Ludvigsson (2019). "Mortality in IgA Nephropathy: A Nationwide Population-Based Cohort Study." <u>J Am Soc Nephrol</u> **30**(5): 866-876.
- KDIGO (2012). "KDIGO Clinical Practice Guideline for Glomerulonephritis." <u>Kidney International Supplements</u> **2**(2): 139-274.
- Kiryluk, K., Y. Li, F. Scolari, S. Sanna-Cherchi, M. Choi, M. Verbitsky, D. Fasel, S. Lata, S. Prakash, S. Shapiro, C. Fischman, H. J. Snyder, G. Appel, C. Izzi, B. F. Viola, N. Dallera, L. Del Vecchio, C. Barlassina, E. Salvi, F. E. Bertinetto, A. Amoroso, S. Savoldi, M. Rocchietti, A. Amore, L. Peruzzi, R. Coppo, M. Salvadori, P. Ravani, R. Magistroni, G. M. Ghiggeri, G. Caridi, M. Bodria, F. Lugani, L. Allegri, M. Delsante, M. Maiorana, A. Magnano, G. Frasca, E. Boer, G. Boscutti, C. Ponticelli, R. Mignani, C. Marcantoni, D. Di Landro, D. Santoro, A. Pani, R. Polci, S. Feriozzi, S. Chicca, M. Galliani, M. Gigante, L. Gesualdo, P. Zamboli, G. G. Battaglia, M. Garozzo, D. Maixnerova, V. Tesar, F. Eitner, T. Rauen, J. Floege, T. Kovacs, J. Nagy, K. Mucha, L. Paczek, M. Zaniew, M. Mizerska-Wasiak, M. Roszkowska-Blaim, K. Pawlaczyk, D. Gale, J. Barratt, L. Thibaudin, F. Berthoux, G. Canaud, A. Boland, M. Metzger, U. Panzer, H. Suzuki, S. Goto, I. Narita, Y. Caliskan, J. Xie, P. Hou, N. Chen, H. Zhang, R. J. Wyatt, J. Novak, B. A. Julian, J. Feehally, B. Stengel, D. Cusi, R. P. Lifton and A. G. Gharavi (2014). "Discovery of new risk loci for IgA nephropathy implicates genes involved in immunity against intestinal pathogens." Nat Genet 46(11): 1187-1196.
- Kiryluk, K., Z. Moldoveanu, J. T. Sanders, T. M. Eison, H. Suzuki, B. A. Julian, J. Novak, A. G. Gharavi and R. J. Wyatt (2011). "Aberrant glycosylation of IgA1 is inherited in both pediatric IgA nephropathy and Henoch-Schonlein purpura nephritis." <u>Kidney Int</u> **80**(1): 79-87.
- Kiryluk, K. and J. Novak (2014). "The genetics and immunobiology of IgA nephropathy." <u>The Journal of Clinical Investigation</u> **124**(6): 2325-2332.

- Kiryluk, K., J. Novak and A. G. Gharavi (2013). "Pathogenesis of immunoglobulin A nephropathy: recent insight from genetic studies." <u>Annual review of medicine</u> **64**: 339-356.
- Knoppova, B., C. Reily, N. Maillard, D. V. Rizk, Z. Moldoveanu, J. Mestecky, M. Raska, M. B. Renfrow, B. A. Julian and J. Novak (2016). "The Origin and Activities of IgA1-Containing Immune Complexes in IgA Nephropathy." <u>Front Immunol</u> 7: 117.
- Lai, K. N., S. C. Tang, F. P. Schena, J. Novak, Y. Tomino, A. B. Fogo and R. J. Glassock (2016). "IgA nephropathy." <u>Nat Rev Dis Primers</u> **2**: 16001.
- Levey, A. S., L. A. Stevens, C. H. Schmid, Y. L. Zhang, A. F. Castro, 3rd, H. I. Feldman, J. W. Kusek, P. Eggers, F. Van Lente, T. Greene, J. Coresh and E. P. I. Ckd (2009). "A new equation to estimate glomerular filtration rate." <u>Ann Intern Med</u> **150**(9): 604-612.
- Louis, A. G., S. Agrawal and S. Gupta (2016). "Analysis of subsets of B cells, Breg, CD4Treg and CD8Treg cells in adult patients with primary selective IgM deficiency." <u>Am J Clin Exp Immunol</u> **5**(1): 21-32.
- Louis, A. G. and S. Gupta (2014). "Primary selective IgM deficiency: an ignored immunodeficiency." Clin Rev Allergy Immunol 46(2): 104-111.
- Lv, J., H. Zhang, M. G. Wong, M. J. Jardine, M. Hladunewich, V. Jha, H. Monaghan, M. Zhao, S. Barbour, H. Reich, D. Cattran, R. Glassock, A. Levin, D. Wheeler, M. Woodward, L. Billot, T. M. Chan, Z. H. Liu, D. W. Johnson, A. Cass, J. Feehally, J. Floege, G. Remuzzi, Y. Wu, R. Agarwal, H. Y. Wang and V. Perkovic (2017). "Effect of Oral Methylprednisolone on Clinical Outcomes in Patients With IgA Nephropathy: The TESTING Randomized Clinical Trial." <u>Jama</u> **318**(5): 432-442.
- Mestecky, J., J. Novak, Z. Moldoveanu and M. Raska (2016). "IgA nephropathy enigma." <u>Clin</u> Immunol **172**: 72-77.
- Mestecky, J., M. Raska, B. A. Julian, A. G. Gharavi, M. B. Renfrow, Z. Moldoveanu, L. Novak, K. Matousovic and J. Novak (2013). "IgA nephropathy: molecular mechanisms of the disease." Annu Rev Pathol 8: 217-240.
- Muto, M., B. Manfroi, H. Suzuki, K. Joh, M. Nagai, S. Wakai, C. Righini, M. Maiguma, S. Izui, Y. Tomino, B. Huard and Y. Suzuki (2017). "Toll-Like Receptor 9 Stimulation Induces Aberrant Expression of a Proliferation-Inducing Ligand by Tonsillar Germinal Center B Cells in IgA Nephropathy." J Am Soc Nephrol **28**(4): 1227-1238.
- Myette, J. R., T. Kano, H. Suzuki, S. E. Sloan, K. J. Szretter, B. Ramakrishnan, H. Adari, K. D. Deotale, F. Engler, Z. Shriver, A. M. Wollacott, Y. Suzuki and B. J. G. Pereira (2019). "A Proliferation Inducing Ligand (APRIL) targeted antibody is a safe and effective treatment of murine IgA nephropathy." <u>Kidney International</u> **96**(1): 104-116.
- Nam, K. H., J. H. Kie, M. J. Lee, T. I. Chang, E. W. Kang, D. W. Kim, B. J. Lim, J. T. Park, Y. E. Kwon, Y. L. Kim, K. S. Park, S. Y. An, H. J. Oh, T. H. Yoo, S. W. Kang, K. H. Choi, H. J. Jeong, D. S. Han and S. H. Han (2014). "Optimal proteinuria target for renoprotection in patients with IgA nephropathy." <u>PLoS One</u> **9**(7): e101935.

Pozzi, C., S. Andrulli, L. Del Vecchio, P. Melis, G. B. Fogazzi, P. Altieri, C. Ponticelli and F. Locatelli (2004). "Corticosteroid effectiveness in IgA nephropathy: long-term results of a randomized, controlled trial." J Am Soc Nephrol **15**(1): 157-163.

Radhakrishnan, J. and D. C. Cattran (2012). "The KDIGO practice guideline on glomerulonephritis: reading between the (guide)lines--application to the individual patient." Kidney Int 82(8): 840-856.

Rauen, T., F. Eitner, C. Fitzner, C. Sommerer, M. Zeier, B. Otte, U. Panzer, H. Peters, U. Benck, P. R. Mertens, U. Kuhlmann, O. Witzke, O. Gross, V. Vielhauer, J. F. Mann, R. D. Hilgers and J. Floege (2015). "Intensive Supportive Care plus Immunosuppression in IgA Nephropathy." <u>N Engl J Med</u> **373**(23): 2225-2236.

Reich, H. N., S. Troyanov, J. W. Scholey and D. C. Cattran (2007). "Remission of proteinuria improves prognosis in IgA nephropathy." J Am Soc Nephrol 18(12): 3177-3183.

Rodrigues, J. C., M. Haas and H. N. Reich (2017). "IgA Nephropathy." <u>Clinical Journal of the American Society of Nephrology</u> **12**(4): 677-686.

Schena, F. P. and I. Nistor (2018). "Epidemiology of IgA Nephropathy: A Global Perspective." <u>Semin Nephrol</u> **38**(5): 435-442.

Tesar, V., S. Troyanov, S. Bellur, J. C. Verhave, H. T. Cook, J. Feehally, I. S. Roberts, D. Cattran and R. Coppo (2015). "Corticosteroids in IgA Nephropathy: A Retrospective Analysis from the VALIGA Study." <u>J Am Soc Nephrol</u> **26**(9): 2248-2258.

Thompson, A., K. Carroll, L. A. Inker, J. Floege, V. Perkovic, S. Boyer-Suavet, R. W. Major, J. I. Schimpf, J. Barratt, D. C. Cattran, B. S. Gillespie, A. Kausz, A. W. Mercer, H. N. Reich, B. H. Rovin, M. West and P. H. Nachman (2019). "Proteinuria Reduction as a Surrogate End Point in Trials of IgA Nephropathy." <u>Clinical Journal of the American Society of Nephrology</u> **14**(3): 469-481.

Trimarchi, H., J. Barratt, D. C. Cattran, H. T. Cook, R. Coppo, M. Haas, Z. H. Liu, I. S. Roberts, Y. Yuzawa, H. Zhang and J. Feehally (2017). "Oxford Classification of IgA nephropathy 2016: an update from the IgA Nephropathy Classification Working Group." <u>Kidney Int</u> **91**(5): 1014-1021.

Varfolomeev, E., F. Kischkel, F. Martin, D. Seshasayee, H. Wang, D. Lawrence, C. Olsson, L. Tom, S. Erickson, D. French, P. Schow, I. S. Grewal and A. Ashkenazi (2004). "APRIL-deficient mice have normal immune system development." <u>Mol Cell Biol</u> **24**(3): 997-1006.

Working Group of the International Ig, A. N. N., S. the Renal Pathology, D. C. Cattran, R. Coppo, H. T. Cook, J. Feehally, I. S. Roberts, S. Troyanov, C. E. Alpers, A. Amore, J. Barratt, F. Berthoux, S. Bonsib, J. A. Bruijn, V. D'Agati, G. D'Amico, S. Emancipator, F. Emma, F. Ferrario, F. C. Fervenza, S. Florquin, A. Fogo, C. C. Geddes, H. J. Groene, M. Haas, A. M. Herzenberg, P. A. Hill, R. J. Hogg, S. I. Hsu, J. C. Jennette, K. Joh, B. A. Julian, T. Kawamura, F. M. Lai, C. B. Leung, L. S. Li, P. K. Li, Z. H. Liu, B. Mackinnon, S. Mezzano, F. P. Schena, Y. Tomino, P. D. Walker, H. Wang, J. J. Weening, N. Yoshikawa and H. Zhang (2009). "The

Oxford classification of IgA nephropathy: rationale, clinicopathological correlations, and classification." <u>Kidney Int</u> **76**(5): 534-545.

Wyatt, R. J. and B. A. Julian (2013). "IgA nephropathy." N Engl J Med 368(25): 2402-2414.

Yazdani, R., G. Azizi, H. Abolhassani and A. Aghamohammadi (2017). "Selective IgA Deficiency: Epidemiology, Pathogenesis, Clinical Phenotype, Diagnosis, Prognosis and Management." <u>Scand J Immunol</u> **85**(1): 3-12.

Yel, L., S. Ramanuja and S. Gupta (2009). "Clinical and immunological features in IgM deficiency." Int Arch Allergy Immunol 150(3): 291-298.

Zhai, Y. L., L. Zhu, S. F. Shi, L. J. Liu, J. C. Lv and H. Zhang (2016). "Increased APRIL Expression Induces IgA1 Aberrant Glycosylation in IgA Nephropathy." <u>Medicine (Baltimore)</u> **95**(11): e3099.

Zhao, N., P. Hou, J. Lv, Z. Moldoveanu, Y. Li, K. Kiryluk, A. G. Gharavi, J. Novak and H. Zhang (2012). "The level of galactose-deficient IgA1 in the sera of patients with IgA nephropathy is associated with disease progression." <u>Kidney Int</u> **82**(7): 790-796.